CLINICAL TRIAL: NCT06607471
Title: Multimodal and Multidisciplinary Approach to Optimize Diagnostic, Prognostic, and Therapeutic Management of Patients with Non-ischemic Cardiomyopathies and Arrhythmogenic-inflammatory Phenotypes: a Multicenter, Observational, Retrospective and Prospective Registry Study.
Acronym: AINICM
Status: Recruiting | Type: Observational
Sponsor: Scientific Institute San Raffaele (Other)
Responsible Party: Principal Investigator, Giovanni Peretto, MD, Principal Investigator, Scientific Institute San Raffaele
Other Study IDs: AINICM
Record Dates: First submitted 2024-09-07; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Non-ischemic Cardiomyopathy; Dilated Cardiomyopathy (DCM); Hypertrophic Cardiomyopathy (HCM); Restrictive Cardiomyopathy; Arrhythmogenic Cardiomyopathy (AC, ARVD/C); Left Ventricular Noncompaction; Arrhythmogenic Mitral Valve Prolapse; Peripartum Cardiomyopathy; Anderson-Fabry Disease; Arrhythmic and Inflammatory Non-ischemic Cardiomyopathy; Inflammatory (Non-Arrhythmic) Non-ischemic Cardiomyopathy; Nonischemic Cardiomyopathy Sensu Strictu (Non-inflammatory, Non-arrhythmic); Major Ventricular Arrhythmias, I.e. Sustained Ventricular Tachycardia, Ventricular Fibrillation, or Appropriate Therapy of Cardiac Device (defibrillators); Overlapping Phenotype; Undefined Phenotypes
Keywords: Arrhythmogenic cardiomyopathy; Adverse event; Anderson-Fabry disease; Arrhythmic and Inflammatory Non-ischemic cardiomyopathy; Arrhythmogenic mitral valve prolapse; Anti tachycardia pacing; Bradiarrhythmias; Cardiac magnetic resonance; Cardiac resynchronization therapy with defibrillator; Computed tomography; Development Safety Update Report; Ethics Committee; Electroanatomical map; Electrocardiogram; Endomyocardial biopsy; Good Clinical Practice; Hypertrophic cardiomyopathy; Implantable cardioverter defibrillator; Informed Consent Form; International Conference on Harmonization; Immunomodulatory therapy; Late gadolinium enhancement; Left ventricular ejection fraction; Left ventricular noncompaction; Last Visit of Last Subject; Myocardial inflammation; Non-ischemic cardiomyopathies; Positron emission tomography; Pacemaker; Peripartum cardiomyopathy; Premature ventricular complexes; Serious Adverse Event; Supraventricular arrhythmias; Ventricular arrhythmias; Ventricular fibrillation; Ventricular tachycardia (sustained); sudden cardiac death
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Restrictive; Arrhythmogenic Right Ventricular Dysplasia; Peripartum Cardiomyopathy; Fabry Disease; Ventricular Fibrillation; Myocarditis; Ventricular Premature Complexes; Tachycardia, Ventricular; Death, Sudden, Cardiac | interventions — Equipment and Supplies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Biospecimen Retention: Samples With DNA — It includes circulating, tissue and biomarkers. as well as genetic, transcriptomic, proteomic, metabolic, epigenetic markers.
  Undefined a-priori. Will be considered in clinically-indicated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Arrhythmic and Inflammatory (AINICM): The AINICM group will include presentation with ventricular fibrillation (VF), either sustained or non-sustained ventricular tachycardia (VT; NSVT), frequent premature ventricular complexes (PVC), supraventricular arrhythmias (SVA) and bradyarrhythmias (BA).
  The arrhythmogenic and the inflammatory non-ischemic cardiomyopathies (AINICM) will be characterized by means of a multimodal diagnostic workup, which is a combination ofgenetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry.
  Interventions: Other: Support treatment, cardiac medical treatment, aetiology-specific treatment, device implant, arrhythmia ablation
- Non-arrhythmic and inflammatory (INICM): The inflammatory component will be diagnosed by means of a multidisciplinary workup (i.e. EMB, PET).
  Interventions: Other: Support treatment, cardiac medical treatment, aetiology-specific treatment
- Arrhythmic and Non-inflammatory (ANICM): The arrhythmic component will be diagnosed by means of a multidisciplinary work-up (i.e. SAECG, Arrhythmia monitoring, Stress test, CT scan, EAM, Electrophysiological test)
  Interventions: Other: Support treatment, cardiac medical treatment, aetiology-specific treatment, device implant, arrhythmia ablation
- Non-arrhythmic and Non-inflammatory (NICM): NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
  Interventions: Other: Support treatment, cardiac medical treatment, aetiology-specific treatment

INTERVENTIONS:
Other: Support treatment, cardiac medical treatment, aetiology-specific treatment, device implant, arrhythmia ablation — Treatment will be patient-tailored, integrating international guidelines recommendation and the experience of the center where enrollment takes place.
  Groups: Arrhythmic and Inflammatory (AINICM); Arrhythmic and Non-inflammatory (ANICM)
Other: Support treatment, cardiac medical treatment, aetiology-specific treatment — Treatment will be patient-tailored, integrating international guidelines recommendation and the experience of the center where enrollment takes place.
  Groups: Non-arrhythmic and Non-inflammatory (NICM); Non-arrhythmic and inflammatory (INICM)

SUMMARY:
Non-ischemic cardiomyopathies (NICM) represent a heterogeneous group of pathologies characterized by absence of obstructive disease of the epicardial coronary vessels and distinct structural and functional changes of the myocardium. The main identified forms include dilated cardiomyopathy (DCM), hypertrophic cardiomyopathy (HCM), restrictive cardiomyopathy (RCM), and arrhythmogenic cardiomyopathy proper (ACM). More recently, further forms of cardiomyopathy have been described, less common and not uniquely classifiable, including: uncompressed myocardium (LVNC), peripartum cardiomyopathy (PPCM), structural correlates of arrhythmogenic mitral valve prolapse (AMVP), Anderson-Fabry disease (AFD), NICM associated with multi- system neuromuscular or autoimmune diseases, lysosomal diseases, glycogenosis, mitochondrial cytopathies and canal diseases with structural substrates. Finally, there are "overlap" forms, characterized by the sharing in the same subject of characteristic aspects of two or more of the above- mentioned diseases; and of the "undefined" forms, which to date do not reach the diagnostic criteria for any of the above-mentioned diseases.

To the best of current knowledge, there are two points discovered in scientific research, namely the description of the arrhythmogenic and "inflammatory" phenotypes in a broad sense, which are summarized here with the acronym AINICM. In detail:

1. Arrhythmic manifestations account for the arrhythmogenic component of AINICM, which is not limited to ACM proper. In fact, most of the above diseases have a non-arrhythmic clinical presentation and a prevailing tendency to evolve towards a picture of cardiovascular decompensation. Although sudden arrhythmic death has been described throughout the spectrum of AINICM, early arrhythmic manifestations of such diseases have an unknown prevalence, an uncertain association with different disease genotypes and phenotypes, and still uncertain predictivity of long-term arrhythmic risk. At the same time, optimal diagnostic and therapeutic pathways in arrhythmias associated with AINICM are still being studied.
2. Myocardial inflammation (M-Infl) accounts for the inflammatory component of AINICM, and has recently been described in association with many AINICM on a genetic basis, including undefined and arrhythmic forms. The data is of high interest not only in the diagnostic, but also in prognostic and therapeutic field. In fact, on the one hand the presence of M-Infl seems to have a physio- pathological role in AINICM; on the other, as already known in myocarditis, the optimal therapeutic paths of arrhythmias may differ in patients with and without M-Infl; in particular, also in the light of the preliminary data available in adult and paediatric AINICM, the inflammatory forms are expected to respond better to immunosuppressive therapy, the arrhythmogenic ones to an ablative therapy with frequent need of implantation of cardiac devices.

Based on the clinical presentation, NICM patients will be divided into arrhythmic (AINICM) and non-arrhythmic patients as study and control groups , respectively. The AINICM group will include presentation with ventricular fibrillation (VF), either sustained or non-sustained ventricular tachycardia (VT; NSVT), frequent premature ventricular complexes (PVC), supraventricular arrhythmias (SVA) and bradyarrhythmias (BA). Clinical presentations other than arrhythmic, including chest pain and heart failure, will define the control group. In parallel, as shown in Figure 1, patients with any evidence of M-Infl will be compared with those showing no signs of M-Infl.

DETAILED DESCRIPTION:
This study aims to collect clinical data of both retrospective and prospective patients with suspected or proven NICMs in a registry. The scope of the registry is to answer multiple unsolved questions in the field of AINICM as described below:

1. Improving the diagnostic workup. While genetic test and cardiac magnetic resonance (CMR) constitute the gold standard dagnostic techniques for NICM, it is known that; A) the yield of genetic test is low in NICM; B) the diagnostic performance of CMR may be limited in AINICM, because of cardiac device-related artifacts and/or irregular heartbeat. In this setting, alternative diagnostic techniques, namely computed tomography (CT) scan, positron emission tomography (PET), electroanatomical map (EAM) and endomyocardial biopsy (EMB) may be clinically helpful, as recommended for the investigation of many arrhythmogenic substrates.
2. Identifying disease-specific signatures. Genotype-phenoype associations are expected to benefit from a multimodal and multiparametric approach, in order to allow etiology-specific features in AINICM. Most of the current signatures are limited to combined genotype-CMR studies. Signatures would likely benefit from implementing additional parameters, including arrhythmia features and myocadial inflammatory status.
3. Working our models for risk prediction. Outcomes and arrhythmic risk stratification remain uncertain for most NICM. Based on an advanced multimodal workup, multiparametric risk scores may be created and subsequenlty validated, in order to predict the arrhythmic risk of specific cardiomyopathies. This would improve and refine the scores currently available for a limited number of NICM, such as HCM, classic right ventricular ACM, or cardiomyopathies secondary to LMNA gene mutation. Parameters from clinical arrhythmology and cardiac electrophysiology, as well as those related to inflammation, may improve the current status of the art about risk prediction.
4. Tailoring treatment strategies. A multimodal (i.e. by use of multiple diagnostic techniques) and multidisciplinary (i.e. by means of a team of cardiac electrophysiologists, cardiologists, radiologists, geneticists, immunologists, cardiac pathologists, pediatricians) model may help improving therapeutic strategies in AINICM, as already demonstrated in myocarditis. In detail, treatment options will include guideline-directed cardiological treatment, implantable cardiac devices, antiarrhythmic drugs, immunomodulating agents and catheter ablation of arrhythmias. In this setting, the coordinating center is an internationally recognized third-level referral center for the management of ventricular arrhythmias, and already has advanced facilities, including a dedicated multidisciplinary disease unit for myocarditis and inflammatory cardiomyopathies. In this setting, preliminary evidence suggests a potential benefit from targeting M-Infl even in NICM and AINICM.
5. Allowing direct comparison among specific NICM subgroups. Extensive inclusion criteria, allowing the entry of all NICM in a common registry with homogeneous variables would enable the direct comparison of different AINICM types, by means of multiparametric and multimodal characterization, for the first time including both the electrophysiological and inflammatory viewpoints. This is expected to significantly advance the status of knowledge in the field of NICM.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent. For pediatric patients, consent will be obtained by parents, according to the laws applicable in each of the participating countries.
* Clinical suspicion of NICM, and/or proven diagnosis of any NICM and/or genotype consistent with any NICM.

NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.

Exclusion Criteria:

* Absent informed consent.
* Proven diagnosis of cardiac disease alternative to NICM.
* Lack of diagnostic workup suitable for diagnosing NICM, detecting arrhythmias, or detecting M-Infl.
* For patients retrospectively enrolled: lack of active status of follow-up at the enrolling center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an international registry. Enrolment of NICM patients will be performed without restrictions concerning age, gender, ethnicity, social, political, or economical status. Both inpatients and outpatients will be suitable for enrollment. Beyond clinically suspected or proven NICMs, genotype-positive familial cases will be enrolled. The expected sample size is 150000, of whom 5000 will be enrolled at San Raffaele Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 15000 (Estimated)
Dates: Start 2018-01-30 (Actual); Primary Completion 2035-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in DCM | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in DCM | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in DCM | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in DCM | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in DCM | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in DCM | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in DCM | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in HCM | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in HCM | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in HCM | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in HCM | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in HCM | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in HCM | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in HCM | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in RCM | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in RCM | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in RCM | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in RCM | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in RCM | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in RCM | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in RCM | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in ACM | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in ACM | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in ACM | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in ACM | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in ACM | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in ACM | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in ACM | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in LVNC | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in LVNC | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in LVNC | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in LVNC | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in LVNC | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in LVNC | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in LVNC | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AMVP | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AMVP | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AMVP | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AMVP | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AMVP | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AMVP | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AMVP | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in PPCM | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in PPCM | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in PPCM | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in PPCM | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in PPCM | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in PPCM | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in PPCM | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AFD | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AFD | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AFD | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AFD | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AFD | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AFD | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in AFD | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in storage and dysmetabolic diseases | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in storage and dysmetabolic diseases | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in storage and dysmetabolic diseases | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in storage and dysmetabolic diseases | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in storage and dysmetabolic diseases | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in storage and dysmetabolic diseases | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in storage and dysmetabolic diseases | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in mitochondrial diseases | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in mitochondrial diseases | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in mitochondrial diseases | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in mitochondrial diseases | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in mitochondrial diseases | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in mitochondrial diseases | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in mitochondrial diseases | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in channelopathies with structural changes | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in channelopathies with structural changes | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in channelopathies with structural changes | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in channelopathies with structural changes | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in channelopathies with structural changes | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in channelopathies with structural changes | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in channelopathies with structural changes | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in overlapping phenotypes | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in overlapping phenotypes | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in overlapping phenotypes | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in overlapping phenotypes | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in overlapping phenotypes | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in overlapping phenotypes | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in overlapping phenotypes | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in undefined phenotypes | At baseline
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in undefined phenotypes | At year 5
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in undefined phenotypes | At year 10
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in undefined phenotypes | At year 15
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in undefined phenotypes | At year 20
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in undefined phenotypes | At year 25
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of diagnostic accuracy (in terms of true/false positive/negative rates) amongst different diagnostic techniques in undefined phenotypes | At year 30
  Diagnostic concordance in terms of sensitivity, specificity, positive predictive value, negative predictive value
Assessment of prevalence of M-Inf in DCM, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in DCM, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in DCM, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in DCM, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in DCM, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in DCM, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in DCM, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in HCM, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in HCM, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in HCM, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in HCM, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in HCM, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in HCM, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in HCM, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in RCM, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in RCM, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in RCM, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in RCM, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in RCM, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in RCM, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in RCM, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in ACM, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in ACM, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in ACM, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in ACM, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in ACM, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in ACM, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in ACM, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in LVNC, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in LVNC, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in LVNC, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in LVNC, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in LVNC, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in LVNC, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in LVNC, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AMVP, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AMVP, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AMVP, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AMVP, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AMVP, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AMVP, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AMVP, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in PPCM, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in PPCM, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in PPCM, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in PPCM, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in PPCM, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in PPCM, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in PPCM, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AFD, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AFD, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AFD, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AFD, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AFD, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AFD, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in AFD, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in mitochondrial diseases, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in channelopathies with structural changes, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in overlapping phenotypes, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in overlapping phenotypes, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in overlapping phenotypes, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in overlapping phenotypes, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in overlapping phenotypes, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in overlapping phenotypes, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in overlapping phenotypes, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in undefined phenotypes, as defined by multimodal diagnostic workup | At baseline
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in undefined phenotypes, as defined by multimodal diagnostic workup | At year 5
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in undefined phenotypes, as defined by multimodal diagnostic workup | At year 10
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in undefined phenotypes, as defined by multimodal diagnostic workup | At year 15
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in undefined phenotypes, as defined by multimodal diagnostic workup | At year 20
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in undefined phenotypes, as defined by multimodal diagnostic workup | At year 25
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of M-Inf in undefined phenotypes, as defined by multimodal diagnostic workup | At year 30
  Multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in DCM, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in DCM, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in DCM, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in DCM, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in DCM, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in DCM, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in DCM, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in HCM, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in HCM, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in HCM, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in HCM, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in HCM, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in HCM, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in HCM, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in RCM, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in RCM, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in RCM, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in RCM, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in RCM, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in RCM, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in RCM, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in ACM, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in ACM, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in ACM, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in ACM, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in ACM, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in ACM, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in ACM, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in LVNC, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in LVNC, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in LVNC, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in LVNC, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in LVNC, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in LVNC, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in LVNC, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AMVP, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AMVP, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AMVP, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AMVP, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AMVP, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AMVP, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AMVP, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in PPCM, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in PPCM, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in PPCM, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in PPCM, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in PPCM, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in PPCM, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in PPCM, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AFD, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AFD, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AFD, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AFD, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AFD, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AFD, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in AFD, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in storage and dysmetabolic diseases, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in mitochondrial diseases, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in mitochondrial diseases, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in channelopathies with structural changes, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in channelopathies with structural changes, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of arrhythmogenic substrates in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of overlapping phenotypes, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of overlapping phenotypes, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of overlapping phenotypes, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of overlapping phenotypes, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of overlapping phenotypes, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of overlapping phenotypes, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of overlapping phenotypes, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of undefined phenotypes, as defined by multimodal diagnostic workup | At baseline
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of undefined phenotypes, as defined by multimodal diagnostic workup | At year 5
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of undefined phenotypes, as defined by multimodal diagnostic workup | At year 10
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of undefined phenotypes, as defined by multimodal diagnostic workup | At year 15
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of undefined phenotypes, as defined by multimodal diagnostic workup | At year 20
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of undefined phenotypes, as defined by multimodal diagnostic workup | At year 25
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Assessment of prevalence of undefined phenotypes, as defined by multimodal diagnostic workup | At year 30
  The multimodal diagnostic workup is a combination of genetic tests, different techniques of cardiac imaging, laboratory tests and biomarkers, histology, and electrophysiological tools, collecting all the clinical variables in a registry
Identification of DCM-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of DCM-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of DCM-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of DCM-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of DCM-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of DCM-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of DCM-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of HCM-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of HCM-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of HCM-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of HCM-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of HCM-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of HCM-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of HCM-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of RCM-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of RCM-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of RCM-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of RCM-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of RCM-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of RCM-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of RCM-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of ACM-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of ACM-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of ACM-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of ACM-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of ACM-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of ACM-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of ACM-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of LVNC-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of LVNC-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of LVNC-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of LVNC-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of LVNC-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of LVNC-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of LVNC-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AMVP-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AMVP-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AMVP-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AMVP-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AMVP-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AMVP-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AMVP-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of PPCM-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of PPCM-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of PPCM-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of PPCM-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of PPCM-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of PPCM-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of PPCM-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AFD-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AFD-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AFD-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AFD-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AFD-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AFD-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of AFD-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of storage and dysmetabolic diseases-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of storage and dysmetabolic diseases-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of storage and dysmetabolic diseases-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of storage and dysmetabolic diseases-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of storage and dysmetabolic diseases-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of storage and dysmetabolic diseases-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of storage and dysmetabolic diseases-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of mitochondrial diseases-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of mitochondrial diseases-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of mitochondrial diseases-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of mitochondrial diseases-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of mitochondrial diseases-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of mitochondrial diseases-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of mitochondrial diseases-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of channelopathies with structural changes-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of channelopathies with structural changes-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of channelopathies with structural changes-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of channelopathies with structural changes-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of channelopathies with structural changes-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of channelopathies with structural changes-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of channelopathies with structural changes-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of overlapping phenotypes-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of overlapping phenotypes-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of overlapping phenotypes-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of overlapping phenotypes-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of overlapping phenotypes-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of overlapping phenotypes-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of overlapping phenotypes-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of undefined phenotypes-specific signatures | At baseline
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of undefined phenotypes-specific signatures | At year 5
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of undefined phenotypes-specific signatures | At year 10
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of undefined phenotypes-specific signatures | At year 15
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of undefined phenotypes-specific signatures | At year 20
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of undefined phenotypes-specific signatures | At year 25
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Identification of undefined phenotypes-specific signatures | At year 30
  Identification of disease-specific signatures of diagnosis, etiology, genotype, clinical presentation, arrhythmia type, myocardial inflammation, outcomes, and response to treatment.
Differences in incidence of major events during follow-up in different NICMs | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearanc e/recurrence of M-Infl.
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Differences in incidence of major events during follow-up in different NICMs | At year 5
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearanc e/recurrence of M-Infl.
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Differences in incidence of major events during follow-up in different NICMs | At year 10
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearanc e/recurrence of M-Infl.
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Differences in incidence of major events during follow-up in different NICMs | At year 15
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearanc e/recurrence of M-Infl.
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Differences in incidence of major events during follow-up in different NICMs | At year 20
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearanc e/recurrence of M-Infl.
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Differences in incidence of major events during follow-up in different NICMs | At year 25
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearanc e/recurrence of M-Infl.
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Differences in incidence of major events during follow-up in different NICMs | At year 30
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearanc e/recurrence of M-Infl.
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Occurrence of major cardiac events in DCM | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearanc e/recurrence of M-Infl.
Occurrence of major cardiac events in DCM | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in DCM | At 3 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in DCM | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in DCM | At 15 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in DCM | At 20 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in DCM | At 25 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in DCM | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in HCM | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in HCM | At 3 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in HCM | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in HCM | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in HCM | At 15 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in HCM | At 20 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in HCM | At 25 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in HCM | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in RCM | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in RCM | At 3 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in RCM | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in RCM | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in RCM | At 15 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in RCM | At 20 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in RCM | At 25 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in RCM | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in ACM | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in ACM | At 3 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in ACM | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in ACM | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in ACM | At 15 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in ACM | At 20 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in ACM | At 25 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in ACM | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in LVNC | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in LVNC | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in LVNC | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in LVNC | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in AMVP | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in AMVP | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in AMVP | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in AMVP | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in PPCM | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in PPCM | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in PPCM | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in PPCM | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in AFD | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in AFD | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in AFD | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in AFD | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in storage and dysmetabolic diseases | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in storage and dysmetabolic diseases | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in storage and dysmetabolic diseases | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in storage and dysmetabolic diseases | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in mitochondrial diseases | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in mitochondrial diseases | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in mitochondrial diseases | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in mitochondrial diseases | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in channelopathies with structural changeschannelopathies with structural changes | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in channelopathies with structural changes | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in channelopathies with structural changes | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in channelopathies with structural changes | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in overlapping phenotypes | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in overlapping phenotypes | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in overlapping phenotypes | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in overlapping phenotypes | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in undefined phenotypes | At 1 year
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in undefined phenotypes | At 5 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in undefined phenotypes | At 10 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Occurrence of major cardiac events in undefined phenotypes | At 30 years
  all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in DCM | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in DCM | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in DCM | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in DCM | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in DCM | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in DCM | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in DCM | At 30years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in HCM | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in HCM | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in HCM | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in HCM | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in HCM | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in HCM | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in HCM | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in RCM | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in RCM | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in RCM | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in RCM | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in RCM | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in RCM | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in RCM | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in ACM | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in ACM | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in ACM | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in ACM | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in ACM | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in ACM | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in ACM | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in LVNC | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in LVNC | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in LVNC | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in LVNC | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in LVNC | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in LVNC | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in LVNC | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AMVP | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AMVP | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AMVP | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AMVP | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AMVP | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AMVP | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AMVP | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in PPCM | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in PPCM | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in PPCM | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in PPCM | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in PPCM | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in PPCM | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in PPCM | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AFD | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AFD | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AFD | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AFD | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AFD | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AFD | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in AFD | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in storage and dysmetabolic diseases | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in storage and dysmetabolic diseases | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in storage and dysmetabolic diseases | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in storage and dysmetabolic diseases | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in storage and dysmetabolic diseases | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in storage and dysmetabolic diseases | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in storage and dysmetabolic diseases | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in mitochondrial diseases | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in mitochondrial diseases | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in mitochondrial diseases | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in mitochondrial diseases | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in mitochondrial diseases | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in mitochondrial diseases | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in mitochondrial diseases | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in channelopathies with structural changes | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in channelopathies with structural changes | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in channelopathies with structural changes | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in channelopathies with structural changes | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in channelopathies with structural changes | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in channelopathies with structural changes | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in channelopathies with structural changes | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in overlapping phenotypes | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in overlapping phenotypes | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in overlapping phenotypes | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in overlapping phenotypes | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in overlapping phenotypes | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in overlapping phenotypes | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in overlapping phenotypes | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in undefined phenotypes | At baseline
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in undefined phenotypes | At 5 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in undefined phenotypes | At 10 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in undefined phenotypes | At 15 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in undefined phenotypes | At 20 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in undefined phenotypes | At 25 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.
Evaluation of efficacy of treatment, defined based on the incidence of major events during follow-up in undefined phenotypes | At 30 years
  Real world efficacy (by comparison of outcomes in patients receiving distinct treatment options) and safety profile (complications, side effects) of every therapeutic strategy, either alone or in combination.
  Major events are defined as all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Inf.

SECONDARY OUTCOMES:
Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICM | At baseline
  Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICMs, which include but not limit to DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICM | At 5 years
  Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICMs, which include but not limit to DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICM | At 10 years
  Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICMs, which include but not limit to DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICM | At 15 years
  Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICMs, which include but not limit to DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICM | At 20 years
  Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICMs, which include but not limit to DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICM | At 25 years
  Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICMs, which include but not limit to DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICM | At 30 years
  Prevalence of inflammatory activity (presence; type; quantification; pattern) in NICMs, which include but not limit to DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of inflammatory activity (presence; type; quantification; pattern) in DCM | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in DCM | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in DCM | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in DCM | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in DCM | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in DCM | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in DCM | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in HCM | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in HCM | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in HCM | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in HCM | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in HCM | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in HCM | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in HCM | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in RCM | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in RCM | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in RCM | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in RCM | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in RCM | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in RCM | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in RCM | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in ACM | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in ACM | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in ACM | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in ACM | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in ACM | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in ACM | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in ACM | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in LVNC | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in LVNC | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in LVNC | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in LVNC | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in LVNC | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in LVNC | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in LVNC | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in AMVP | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in AMVP | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in AMVP | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in AMVP | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in AMVP | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in AMVP | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in AMVP | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in PPCM | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in PPCM | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in PPCM | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in PPCM | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in PPCM | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in PPCM | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in PPCM | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in storage and dysmetabolic diseases | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in storage and dysmetabolic diseases | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in storage and dysmetabolic diseases | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in storage and dysmetabolic diseases | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in storage and dysmetabolic diseases | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in storage and dysmetabolic diseases | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in storage and dysmetabolic diseases | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in mitochondrial diseases | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in mitochondrial diseases | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in mitochondrial diseases | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in mitochondrial diseases | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in mitochondrial diseases | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in mitochondrial diseases | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in mitochondrial diseases | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in channelopathies with structural changes | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in channelopathies with structural changes | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in channelopathies with structural changes | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in channelopathies with structural changes | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in channelopathies with structural changes | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in channelopathies with structural changes | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in channelopathies with structural changes | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in overlapping phenotypes | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in overlapping phenotypes | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in overlapping phenotypes | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in overlapping phenotypes | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in overlapping phenotypes | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in overlapping phenotypes | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in overlapping phenotypes | At 30 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in undefined phenotypes | At baseline
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in undefined phenotypes | At 5 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in undefined phenotypes | At 10 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in undefined phenotypes | At 15 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in undefined phenotypes | At 20 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in undefined phenotypes | At 25 years
  presence; type; quantification; pattern
Prevalence of inflammatory activity (presence; type; quantification; pattern) in undefined phenotypes | At 30 years
  presence; type; quantification; pattern
Analysis of correlation between M-Infl and arrhythmia type and ECG features in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between M-Infl and arrhythmia type and ECG features in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between M-Infl and arrhythmia type and ECG features in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between M-Infl and arrhythmia type and ECG features in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between M-Infl and arrhythmia type and ECG features in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between M-Infl and arrhythmia type and ECG features in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between M-Infl and arrhythmia type and ECG features in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between M-Infl and arrhythmia type and ECG features in DCM | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in DCM | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in DCM | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in DCM | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in DCM | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in DCM | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in DCM | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in HCM | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in HCM | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in HCM | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in HCM | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in HCM | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in HCM | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in HCM | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in RCM | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in RCM | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in RCM | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in RCM | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in RCM | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in RCM | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in RCM | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in ACM | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in ACM | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in ACM | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in ACM | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in ACM | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in ACM | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in ACM | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in LVNC | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in LVNC | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in LVNC | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in LVNC | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in LVNC | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in LVNC | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in LVNC | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AMVP | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AMVP | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AMVP | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AMVP | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AMVP | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AMVP | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AMVP | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in PPCM | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in PPCM | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in PPCM | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in PPCM | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in PPCM | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in PPCM | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in PPCM | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AFD | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AFD | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AFD | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AFD | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AFD | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AFD | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in AFD | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in storage and dysmetabolic diseases | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in storage and dysmetabolic diseases | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in storage and dysmetabolic diseases | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in storage and dysmetabolic diseases | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in storage and dysmetabolic diseases | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in storage and dysmetabolic diseases | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in storage and dysmetabolic diseases | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in mitochondrial diseases | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in mitochondrial diseases | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in mitochondrial diseases | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in mitochondrial diseases | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in mitochondrial diseases | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in mitochondrial diseases | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in mitochondrial diseases | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in channelopathies with structural changes | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in channelopathies with structural changes | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in channelopathies with structural changes | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in channelopathies with structural changes | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in channelopathies with structural changes | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in channelopathies with structural changes | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in channelopathies with structural changes | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in overlapping phenotypes | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in overlapping phenotypes | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in overlapping phenotypes | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in overlapping phenotypes | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in overlapping phenotypes | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in overlapping phenotypes | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in overlapping phenotypes | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in undefined phenotypes | At baseline
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in undefined phenotypes | At 5 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in undefined phenotypes | At 10 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in undefined phenotypes | At 15 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in undefined phenotypes | At 20 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in undefined phenotypes | At 25 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between M-Infl and arrhythmia type and ECG features in undefined phenotypes | At 30 years
  correlation between M-Infl and arrhythmia type and ECG features
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, neuromuscular, mitochondrial, toxic, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in DCM | At baseline
  correlation between EMB sampling site and localization of substrate correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in DCM | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in DCM | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in DCM | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in DCM | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in DCM | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in DCM | At 30 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in HCM | At baseline
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in HCM | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in HCM | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in HCM | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in HCM | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in HCM | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in HCM | At 30 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in RCM | At baseline
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in RCM | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in RCM | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in RCM | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in RCM | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in RCM | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in RCM | At 30 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in ACM | At baseline
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in ACM | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in ACM | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in ACM | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in ACM | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in ACM | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in ACM | At 30 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in LVNC | At baseline
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in LVNC | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in LVNC | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in LVNC | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in LVNC | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in LVNC | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in LVNC | At 30 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AMVP | At baseline
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AMVP | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AMVP | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AMVP | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AMVP | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AMVP | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AMVP | At 30 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in PPCM | At baseline
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in PPCM | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in PPCM | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in PPCM | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in PPCM | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in PPCM | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in PPCM | At 30 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AFD | At baseline
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AFD | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AFD | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AFD | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AFD | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AFD | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in AFD | At 30 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in storage and dysmetabolic diseases and mitochondrial diseases | At baseline
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in storage and dysmetabolic diseases and mitochondrial diseases | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in storage and dysmetabolic diseases and mitochondrial diseases | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in storage and dysmetabolic diseases and mitochondrial diseases | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in storage and dysmetabolic diseases and mitochondrial diseases | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in storage and dysmetabolic diseases and mitochondrial diseases | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in storage and dysmetabolic diseases and mitochondrial diseases | At 30 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in channelopathies with structural changes | At baseline
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in channelopathies with structural changes | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in channelopathies with structural changes | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in channelopathies with structural changes | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in channelopathies with structural changes | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in channelopathies with structural changes | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in channelopathies with structural changes | At 30 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in cardiomyopathies associated with systemic, rheumatologic, neuromuscular diseases | At baseline
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in cardiomyopathies associated with systemic, rheumatologic, neuromuscular diseases | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in cardiomyopathies associated with systemic, rheumatologic, neuromuscular diseases | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in cardiomyopathies associated with systemic, rheumatologic, neuromuscular diseases | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in cardiomyopathies associated with systemic, rheumatologic, neuromuscular diseases | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in cardiomyopathies associated with systemic, rheumatologic, neuromuscular diseases | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in cardiomyopathies associated with systemic, rheumatologic, neuromuscular diseases | At 30 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in overlapping and/or undefined phenotypes | At baseline
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in overlapping and/or undefined phenotypes | At 5 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in overlapping and/or undefined phenotypes | At 10 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in overlapping and/or undefined phenotypes | At 15 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in overlapping and/or undefined phenotypes | At 20 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in overlapping and/or undefined phenotypes | At 25 years
  correlation between EMB sampling site and localization of substrate
Analysis of correlation between EMB sampling site and localization of substrate abnormalities at imaging (including substrate-guided EMB or alternative biopsy techniques) in overlapping and/or undefined phenotypes | At 30 years
  correlation between EMB sampling site and localization of substrate
Diagnostic yield of EMB guided by electroanatomical map in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic yield of EMB guided by electroanatomical map in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic yield of EMB guided by electroanatomical map in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic yield of EMB guided by electroanatomical map in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic yield of EMB guided by electroanatomical map in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic yield of EMB guided by electroanatomical map in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic yield of EMB guided by electroanatomical map in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic yield of EMB guided by electroanatomical map in DCM | At baseline
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in DCM | At 5 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in DCM | At 10 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in DCM | At 15 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in DCM | At 20 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in DCM | At 25 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in DCM | At 30 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in HCM | At baseline
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in HCM | At 5 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in HCM | At 10 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in HCM | At 15 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in HCM | At 20 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in HCM | At 25 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in HCM | At 30 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in RCM | At baseline
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in RCM | At 5 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in RCM | At 10 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in RCM | At 15 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in RCM | At 20 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in RCM | At 25 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in RCM | At 30 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in ACM | At baseline
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in ACM | At 5 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in ACM | At 10 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in ACM | At 15 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in ACM | At 20 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in ACM | At 25 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in ACM | At 30 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in LVNC | At baseline
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in LVNC | At 5 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in LVNC | At 10 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in LVNC | At 15 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in LVNC | At 20 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in LVNC | At 25 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in LVNC | At 30 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AMVP | At baseline
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AMVP | At 5 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AMVP | At 10 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AMVP | At 15 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AMVP | At 20 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AMVP | At 25 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AMVP | At 30 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in PPCM | At baseline
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in PPCM | At 5 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in PPCM | At 10 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in PPCM | At 15 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in PPCM | At 20 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in PPCM | At 25 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in PPCM | At 30 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AFD | At baseline
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AFD | At 5 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AFD | At 10 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AFD | At 15 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AFD | At 20 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AFD | At 25 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in AFD | At 30 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in overlapping and/or undefined phenotypes | At baseline
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in overlapping and/or undefined phenotypes | At 5 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in overlapping and/or undefined phenotypes | At 10 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in overlapping and/or undefined phenotypes | At 15 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in overlapping and/or undefined phenotypes | At 20 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in overlapping and/or undefined phenotypes | At 25 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic yield of EMB guided by electroanatomical map in overlapping and/or undefined phenotypes | At 30 years
  Investestigating the role of EMB guided by electroanatomical map in diagnosis
Diagnostic performance of CT scan and/or PET in NICMs, especially when CMR is not feasible | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic performance of CT scan and/or PET in NICMs, especially when CMR is not feasible | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic performance of CT scan and/or PET in NICMs, especially when CMR is not feasible | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic performance of CT scan and/or PET in NICMs, especially when CMR is not feasible | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic performance of CT scan and/or PET in NICMs, especially when CMR is not feasible | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic performance of CT scan and/or PET in NICMs, especially when CMR is not feasible | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic performance of CT scan and/or PET in NICMs, especially when CMR is not feasible | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Comparison between CMR/CT scan/PET/EAM findings (including fusion imaging) and advanced imaging techniques at echocardiogram in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Comparison between CMR/CT scan/PET/EAM findings (including fusion imaging) and advanced imaging techniques at echocardiogram in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Comparison between CMR/CT scan/PET/EAM findings (including fusion imaging) and advanced imaging techniques at echocardiogram in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Comparison between CMR/CT scan/PET/EAM findings (including fusion imaging) and advanced imaging techniques at echocardiogram in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Comparison between CMR/CT scan/PET/EAM findings (including fusion imaging) and advanced imaging techniques at echocardiogram in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Comparison between CMR/CT scan/PET/EAM findings (including fusion imaging) and advanced imaging techniques at echocardiogram in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Comparison between CMR/CT scan/PET/EAM findings (including fusion imaging) and advanced imaging techniques at echocardiogram in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between M-Infl and arrhythmogenic substrates (cause, types, localization, extension, features, outcomes, response to treatment) in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between M-Infl and arrhythmogenic substrates (cause, types, localization, extension, features, outcomes, response to treatment) in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between M-Infl and arrhythmogenic substrates (cause, types, localization, extension, features, outcomes, response to treatment) in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between M-Infl and arrhythmogenic substrates (cause, types, localization, extension, features, outcomes, response to treatment) in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between M-Infl and arrhythmogenic substrates (cause, types, localization, extension, features, outcomes, response to treatment) in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between M-Infl and arrhythmogenic substrates (cause, types, localization, extension, features, outcomes, response to treatment) in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between M-Infl and arrhythmogenic substrates (cause, types, localization, extension, features, outcomes, response to treatment) in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of healing timing of M-Infl in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of healing timing of M-Infl in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of healing timing of M-Infl in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of healing timing of M-Infl in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of healing timing of M-Infl in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of healing timing of M-Infl in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of healing timing of M-Infl in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Association between substrate abnormalities localizations (as assessed by second level imaging techniques) and arrhythmias (type, characteristics and origin site) in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Association between substrate abnormalities localizations (as assessed by second level imaging techniques) and arrhythmias (type, characteristics and origin site) in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Association between substrate abnormalities localizations (as assessed by second level imaging techniques) and arrhythmias (type, characteristics and origin site) in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Association between substrate abnormalities localizations (as assessed by second level imaging techniques) and arrhythmias (type, characteristics and origin site) in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Association between substrate abnormalities localizations (as assessed by second level imaging techniques) and arrhythmias (type, characteristics and origin site) in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Association between substrate abnormalities localizations (as assessed by second level imaging techniques) and arrhythmias (type, characteristics and origin site) in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Association between substrate abnormalities localizations (as assessed by second level imaging techniques) and arrhythmias (type, characteristics and origin site) in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between arrhythmia and inflammation type/features with any other diagnostic exam performed at baseline or during FU | At baseline
  The diagnostic exams mainly include EMB, CMR/CT scan/PET, echocardiogram, stress tests, blood exams, genetic/blood/tissue/cell/molecular/multiomic biomarkers.
  This analysis regards but not limits to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between arrhythmia and inflammation type/features with any other diagnostic exam performed at baseline or during FU | At 5 years
  The diagnostic exams mainly include EMB, CMR/CT scan/PET, echocardiogram, stress tests, blood exams, genetic/blood/tissue/cell/molecular/multiomic biomarkers.
  This analysis regards but not limits to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between arrhythmia and inflammation type/features with any other diagnostic exam performed at baseline or during FU | At 10 years
  The diagnostic exams mainly include EMB, CMR/CT scan/PET, echocardiogram, stress tests, blood exams, genetic/blood/tissue/cell/molecular/multiomic biomarkers.
  This analysis regards but not limits to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between arrhythmia and inflammation type/features with any other diagnostic exam performed at baseline or during FU | At 15 years
  The diagnostic exams mainly include EMB, CMR/CT scan/PET, echocardiogram, stress tests, blood exams, genetic/blood/tissue/cell/molecular/multiomic biomarkers.
  This analysis regards but not limits to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between arrhythmia and inflammation type/features with any other diagnostic exam performed at baseline or during FU | At 20 years
  The diagnostic exams mainly include EMB, CMR/CT scan/PET, echocardiogram, stress tests, blood exams, genetic/blood/tissue/cell/molecular/multiomic biomarkers.
  This analysis regards but not limits to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between arrhythmia and inflammation type/features with any other diagnostic exam performed at baseline or during FU | At 25 years
  The diagnostic exams mainly include EMB, CMR/CT scan/PET, echocardiogram, stress tests, blood exams, genetic/blood/tissue/cell/molecular/multiomic biomarkers.
  This analysis regards but not limits to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of association between arrhythmia and inflammation type/features with any other diagnostic exam performed at baseline or during FU | At 30 years
  The diagnostic exams mainly include EMB, CMR/CT scan/PET, echocardiogram, stress tests, blood exams, genetic/blood/tissue/cell/molecular/multiomic biomarkers.
  This analysis regards but not limits to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of diagnostic accuracy (sensitivity, specificity, positive and negative predictive values) and safety in different diagnostic techniques (EMB, CMR, CT scan, PET; EAM) in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of diagnostic accuracy (sensitivity, specificity, positive and negative predictive values) and safety in different diagnostic techniques (EMB, CMR, CT scan, PET; EAM) in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of diagnostic accuracy (sensitivity, specificity, positive and negative predictive values) and safety in different diagnostic techniques (EMB, CMR, CT scan, PET; EAM) in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of diagnostic accuracy (sensitivity, specificity, positive and negative predictive values) and safety in different diagnostic techniques (EMB, CMR, CT scan, PET; EAM) in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of diagnostic accuracy (sensitivity, specificity, positive and negative predictive values) and safety in different diagnostic techniques (EMB, CMR, CT scan, PET; EAM) in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of diagnostic accuracy (sensitivity, specificity, positive and negative predictive values) and safety in different diagnostic techniques (EMB, CMR, CT scan, PET; EAM) in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of diagnostic accuracy (sensitivity, specificity, positive and negative predictive values) and safety in different diagnostic techniques (EMB, CMR, CT scan, PET; EAM) in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of abnormalities in myocardial structure, function, perfusion, and metabolism in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of abnormalities in myocardial structure, function, perfusion, and metabolism in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of abnormalities in myocardial structure, function, perfusion, and metabolism in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of abnormalities in myocardial structure, function, perfusion, and metabolism in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of abnormalities in myocardial structure, function, perfusion, and metabolism in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of abnormalities in myocardial structure, function, perfusion, and metabolism in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of abnormalities in myocardial structure, function, perfusion, and metabolism in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of non-ischemic myocardial fibrotic scar (presence; type; quantification; pattern; distribution; extension) in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of non-ischemic myocardial fibrotic scar (presence; type; quantification; pattern; distribution; extension) in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of non-ischemic myocardial fibrotic scar (presence; type; quantification; pattern; distribution; extension) in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of non-ischemic myocardial fibrotic scar (presence; type; quantification; pattern; distribution; extension) in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of non-ischemic myocardial fibrotic scar (presence; type; quantification; pattern; distribution; extension) in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of non-ischemic myocardial fibrotic scar (presence; type; quantification; pattern; distribution; extension) in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of non-ischemic myocardial fibrotic scar (presence; type; quantification; pattern; distribution; extension) in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of genetic variants (pathogenic, likely-pahogenic, of unknown significance) in NICMs showing distinct arrhythmic phenotypes, M-Infl and scar patterns | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of genetic variants (pathogenic, likely-pahogenic, of unknown significance) in NICMs showing distinct arrhythmic phenotypes, M-Infl and scar patterns | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of genetic variants (pathogenic, likely-pahogenic, of unknown significance) in NICMs showing distinct arrhythmic phenotypes, M-Infl and scar patterns | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of genetic variants (pathogenic, likely-pahogenic, of unknown significance) in NICMs showing distinct arrhythmic phenotypes, M-Infl and scar patterns | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of genetic variants (pathogenic, likely-pahogenic, of unknown significance) in NICMs showing distinct arrhythmic phenotypes, M-Infl and scar patterns | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of genetic variants (pathogenic, likely-pahogenic, of unknown significance) in NICMs showing distinct arrhythmic phenotypes, M-Infl and scar patterns | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Prevalence of genetic variants (pathogenic, likely-pahogenic, of unknown significance) in NICMs showing distinct arrhythmic phenotypes, M-Infl and scar patterns | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Genotype-phenotype correlations, as assessed by multimodal and multiparametric diagnostic workup in NICMs (i.e. analysis of association between genotypes and distinct imaging/electrocardiographic/inflammatory/laboratory patterns in patients with NICMs) | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Genotype-phenotype correlations, as assessed by multimodal and multiparametric diagnostic workup in NICMs (i.e. analysis of association between genotypes and distinct imaging/electrocardiographic/inflammatory/laboratory patterns in patients with NICMs) | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Genotype-phenotype correlations, as assessed by multimodal and multiparametric diagnostic workup in NICMs (i.e. analysis of association between genotypes and distinct imaging/electrocardiographic/inflammatory/laboratory patterns in patients with NICMs) | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Genotype-phenotype correlations, as assessed by multimodal and multiparametric diagnostic workup in NICMs (i.e. analysis of association between genotypes and distinct imaging/electrocardiographic/inflammatory/laboratory patterns in patients with NICMs) | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Genotype-phenotype correlations, as assessed by multimodal and multiparametric diagnostic workup in NICMs (i.e. analysis of association between genotypes and distinct imaging/electrocardiographic/inflammatory/laboratory patterns in patients with NICMs) | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Genotype-phenotype correlations, as assessed by multimodal and multiparametric diagnostic workup in NICMs (i.e. analysis of association between genotypes and distinct imaging/electrocardiographic/inflammatory/laboratory patterns in patients with NICMs) | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Genotype-phenotype correlations, as assessed by multimodal and multiparametric diagnostic workup in NICMs (i.e. analysis of association between genotypes and distinct imaging/electrocardiographic/inflammatory/laboratory patterns in patients with NICMs) | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of coronary microvascular disease in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of coronary microvascular disease in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of coronary microvascular disease in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of coronary microvascular disease in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of coronary microvascular disease in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of coronary microvascular disease in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of coronary microvascular disease in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of myocardial ischemia in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of myocardial ischemia in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of myocardial ischemia in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of myocardial ischemia in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of myocardial ischemia in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of myocardial ischemia in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of myocardial ischemia in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of autoimmunity in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of autoimmunity in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of autoimmunity in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of autoimmunity in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of autoimmunity in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of autoimmunity in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of autoimmunity in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of any abnormality (genetic, histological, circulating) involving the intercalated disks as known arrhythmogenic players in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of any abnormality (genetic, histological, circulating) involving the intercalated disks as known arrhythmogenic players in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of any abnormality (genetic, histological, circulating) involving the intercalated disks as known arrhythmogenic players in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of any abnormality (genetic, histological, circulating) involving the intercalated disks as known arrhythmogenic players in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of any abnormality (genetic, histological, circulating) involving the intercalated disks as known arrhythmogenic players in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of any abnormality (genetic, histological, circulating) involving the intercalated disks as known arrhythmogenic players in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of any abnormality (genetic, histological, circulating) involving the intercalated disks as known arrhythmogenic players in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of hemodynamic changes in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of hemodynamic changes in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of hemodynamic changes in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of hemodynamic changes in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of hemodynamic changes in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of hemodynamic changes in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of hemodynamic changes in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Multimodal multiparametric imaging investigation of NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Multimodal multiparametric imaging investigation of NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Multimodal multiparametric imaging investigation of NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Multimodal multiparametric imaging investigation of NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Multimodal multiparametric imaging investigation of NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Multimodal multiparametric imaging investigation of NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Multimodal multiparametric imaging investigation of NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of differential diagnosis between NICMs and other cardiac diseases | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of differential diagnosis between NICMs and other cardiac diseases | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of differential diagnosis between NICMs and other cardiac diseases | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of differential diagnosis between NICMs and other cardiac diseases | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of differential diagnosis between NICMs and other cardiac diseases | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of differential diagnosis between NICMs and other cardiac diseases | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Evaluation of differential diagnosis between NICMs and other cardiac diseases | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers of inflammatory stage (acute vs. chronic; active vs. previous) in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers of inflammatory stage (acute vs. chronic; active vs. previous) in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers of inflammatory stage (acute vs. chronic; active vs. previous) in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers of inflammatory stage (acute vs. chronic; active vs. previous) in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers of inflammatory stage (acute vs. chronic; active vs. previous) in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers of inflammatory stage (acute vs. chronic; active vs. previous) in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers of inflammatory stage (acute vs. chronic; active vs. previous) in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between local and systemic/peripheral inflammation in NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between local and systemic/peripheral inflammation in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between local and systemic/peripheral inflammation in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between local and systemic/peripheral inflammation in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between local and systemic/peripheral inflammation in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between local and systemic/peripheral inflammation in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of correlation between local and systemic/peripheral inflammation in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of the concordance/discordance between the diagnostic findings observed in NICMs by means of distinct techniques, namely EMB and imaging (CMR, CT scan, PET, EAM, echocardiogram) | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of the concordance/discordance between the diagnostic findings observed in NICMs by means of distinct techniques, namely EMB and imaging (CMR, CT scan, PET, EAM, echocardiogram) | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of the concordance/discordance between the diagnostic findings observed in NICMs by means of distinct techniques, namely EMB and imaging (CMR, CT scan, PET, EAM, echocardiogram) | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of the concordance/discordance between the diagnostic findings observed in NICMs by means of distinct techniques, namely EMB and imaging (CMR, CT scan, PET, EAM, echocardiogram) | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of the concordance/discordance between the diagnostic findings observed in NICMs by means of distinct techniques, namely EMB and imaging (CMR, CT scan, PET, EAM, echocardiogram) | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of the concordance/discordance between the diagnostic findings observed in NICMs by means of distinct techniques, namely EMB and imaging (CMR, CT scan, PET, EAM, echocardiogram) | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Analysis of the concordance/discordance between the diagnostic findings observed in NICMs by means of distinct techniques, namely EMB and imaging (CMR, CT scan, PET, EAM, echocardiogram) | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Investigation of infectious, toxicologic, and immunologic factors associated with NICMs | At baseline
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Investigation of infectious, toxicologic, and immunologic factors associated with NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Investigation of infectious, toxicologic, and immunologic factors associated with NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Investigation of infectious, toxicologic, and immunologic factors associated with NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Investigation of infectious, toxicologic, and immunologic factors associated with NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Investigation of infectious, toxicologic, and immunologic factors associated with NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Investigation of infectious, toxicologic, and immunologic factors associated with NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic factors with any role in etiology, clinical presentation, diagnosis, prognosis, response to treatment | At baseline
  This will be assessed either in the presence or in the absence of defined NICMs. NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic factors with any role in etiology, clinical presentation, diagnosis, prognosis, response to treatment | At 5 years
  This will be assessed either in the presence or in the absence of defined NICMs. NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic factors with any role in etiology, clinical presentation, diagnosis, prognosis, response to treatment | At 10 years
  This will be assessed either in the presence or in the absence of defined NICMs. NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic factors with any role in etiology, clinical presentation, diagnosis, prognosis, response to treatment | At 15 years
  This will be assessed either in the presence or in the absence of defined NICMs. NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic factors with any role in etiology, clinical presentation, diagnosis, prognosis, response to treatment | At 20 years
  This will be assessed either in the presence or in the absence of defined NICMs. NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic factors with any role in etiology, clinical presentation, diagnosis, prognosis, response to treatment | At 25 years
  This will be assessed either in the presence or in the absence of defined NICMs. NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic factors with any role in etiology, clinical presentation, diagnosis, prognosis, response to treatment | At 30 years
  This will be assessed either in the presence or in the absence of defined NICMs. NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the diagnostic yield of different techniques of arrhythmia monitoring in NICMs | At baseline
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the diagnostic yield of different techniques of arrhythmia monitoring in NICMs | At 5 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the diagnostic yield of different techniques of arrhythmia monitoring in NICMs | At 10 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the diagnostic yield of different techniques of arrhythmia monitoring in NICMs | At 15 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the diagnostic yield of different techniques of arrhythmia monitoring in NICMs | At 20 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the diagnostic yield of different techniques of arrhythmia monitoring in NICMs | At 25 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the diagnostic yield of different techniques of arrhythmia monitoring in NICMs | At 30 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Invasive and noninvasive investigation of arrhythmogenic substrates in NICMs | At baseline
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Invasive and noninvasive investigation of arrhythmogenic substrates in NICMs | At 5 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Invasive and noninvasive investigation of arrhythmogenic substrates in NICMs | At 10 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Invasive and noninvasive investigation of arrhythmogenic substrates in NICMs | At 15 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Invasive and noninvasive investigation of arrhythmogenic substrates in NICMs | At 20 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Invasive and noninvasive investigation of arrhythmogenic substrates in NICMs | At 25 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Invasive and noninvasive investigation of arrhythmogenic substrates in NICMs | At 30 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic value of extracardiac diagnostic techniques in NICMs | At baseline
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic value of extracardiac diagnostic techniques in NICMs | At 5 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic value of extracardiac diagnostic techniques in NICMs | At 10 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic value of extracardiac diagnostic techniques in NICMs | At 15 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic value of extracardiac diagnostic techniques in NICMs | At 20 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic value of extracardiac diagnostic techniques in NICMs | At 25 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Diagnostic value of extracardiac diagnostic techniques in NICMs | At 30 years
  NICMs include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatological/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Occurrence of minor events in DCM | At 1 year
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in DCM | At 3 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in DCM | At 5 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in DCM | At 10 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in DCM | At 15 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in DCM | At 20 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in DCM | At 25 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in DCM | At 30 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in HCM | At 1 year
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in HCM | At 3 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in HCM | At 5 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in HCM | At 10 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in HCM | At 15 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in HCM | At 20 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in HCM | At 25 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in HCM | At 30 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in RCM | At 1 year
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in RCM | At 3 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in RCM | At 5 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in RCM | At 10 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in RCM | At 15 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in RCM | At 20 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence in minor events in RCM | At 25 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in RCM | At 30 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in ACM | At 1 year
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in ACM | At 3 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in ACM | At 5 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in ACM | At 10 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in ACM | At 15 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in ACM | At 20 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in ACM | At 25 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in ACM | At 30 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in distinct cardiomyopathic phenotypes that have been described in some diseases | At 1 year
  left ventricular noncompaction (LVNC), arrhythmogenic mitral valve prolapse (AMVP), peripartum cardiomyopathy (PPCM), Anderson-Fabry disease (AFD), storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases.
  Minor events include non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in distinct cardiomyopathic phenotypes have been described in some diseases | At 5 years
  left ventricular noncompaction (LVNC), arrhythmogenic mitral valve prolapse (AMVP), peripartum cardiomyopathy (PPCM), Anderson-Fabry disease (AFD), storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases.
  Minor events include non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in distinct cardiomyopathic phenotypes that have been described in some diseases | At 10 years
  left ventricular noncompaction (LVNC), arrhythmogenic mitral valve prolapse (AMVP), peripartum cardiomyopathy (PPCM), Anderson-Fabry disease (AFD), storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases.
  Minor events include non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in distinct cardiomyopathic phenotypes that have been described in some diseases | At 30 years
  left ventricular noncompaction (LVNC), arrhythmogenic mitral valve prolapse (AMVP), peripartum cardiomyopathy (PPCM), Anderson-Fabry disease (AFD), storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases.
  Minor events include non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in overlapping and undefined phenotypes | At 1 year
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in overlapping and undefined phenotypes | At 5 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in overlapping and undefined phenotypes | At 10 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Occurrence of minor events in overlapping and undefined phenotypes | At 30 years
  non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Description of the natural history of overall and specific forms of NICM, showing distinct arrhythmic phenotypes, M-Infl and scar patterns. | At 1 year
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Description of the natural history of overall and specific forms of NICM, showing distinct arrhythmic phenotypes, M-Infl and scar patterns. | At 3 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Description of the natural history of overall and specific forms of NICM, showing distinct arrhythmic phenotypes, M-Infl and scar patterns. | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, dysmetabolic, mitochondrial, toxic, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Description of the natural history of overall and specific forms of NICM, showing distinct arrhythmic phenotypes, M-Infl and scar patterns. | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Description of the natural history of overall and specific forms of NICM, showing distinct arrhythmic phenotypes, M-Infl and scar patterns. | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Description of the natural history of overall and specific forms of NICM, showing distinct arrhythmic phenotypes, M-Infl and scar patterns. | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Description of the natural history of overall and specific forms of NICM, showing distinct arrhythmic phenotypes, M-Infl and scar patterns. | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Description of the natural history of overall and specific forms of NICM, showing distinct arrhythmic phenotypes, M-Infl and scar patterns. | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of prognostic genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic biomarkers for NICMs | At 1 year
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of prognostic genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic biomarkers for NICMs | At 3 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of prognostic genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic biomarkers for NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of prognostic genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic biomarkers for NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of prognostic genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic biomarkers for NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of prognostic genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic biomarkers for NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of prognostic genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic biomarkers for NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of prognostic genetic, circulatory, tissue, cellular, metabolic, molecular, immunologic or multiomic biomarkers for NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers associated with treatment response for NICMs | At 1 year
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers associated with treatment response for NICMs | At 3 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers associated with treatment response for NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers associated with treatment response for NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers associated with treatment response for NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers associated with treatment response for NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers associated with treatment response for NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of biomarkers associated with treatment response for NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of cost-effective multimodal and multiparametric risk scores for NICMs | At 1 year
  These risk scores will be aimed but not limit to obtain the maximal capability of discriminating heterogeneous outcomes by means of the minimal number of predictors and/or the minimal number of exams and/or the chepest/safest exams.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of cost-effective multimodal and multiparametric risk scores for NICMs | At 3 years
  These risk scores will be aimed but not limit to obtain the maximal capability of discriminating heterogeneous outcomes by means of the minimal number of predictors and/or the minimal number of exams and/or the chepest/safest exams.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of cost-effective multimodal and multiparametric risk scores for NICMs | At 5 years
  These risk scores will be aimed but not limit to obtain the maximal capability of discriminating heterogeneous outcomes by means of the minimal number of predictors and/or the minimal number of exams and/or the chepest/safest exams.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of cost-effective multimodal and multiparametric risk scores for NICMs | At 10 years
  These risk scores will be aimed but not limit to obtain the maximal capability of discriminating heterogeneous outcomes by means of the minimal number of predictors and/or the minimal number of exams and/or the chepest/safest exams.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of cost-effective multimodal and multiparametric risk scores for NICMs | At 15 years
  These risk scores will be aimed but not limit to obtain the maximal capability of discriminating heterogeneous outcomes by means of the minimal number of predictors and/or the minimal number of exams and/or the chepest/safest exams.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of cost-effective multimodal and multiparametric risk scores for NICMs | At 20 years
  These risk scores will be aimed but not limit to obtain the maximal capability of discriminating heterogeneous outcomes by means of the minimal number of predictors and/or the minimal number of exams and/or the chepest/safest exams.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of cost-effective multimodal and multiparametric risk scores for NICMs | At 25 years
  These risk scores will be aimed but not limit to obtain the maximal capability of discriminating heterogeneous outcomes by means of the minimal number of predictors and/or the minimal number of exams and/or the chepest/safest exams.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of cost-effective multimodal and multiparametric risk scores for NICMs | At 30 years
  These risk scores will be aimed but not limit to obtain the maximal capability of discriminating heterogeneous outcomes by means of the minimal number of predictors and/or the minimal number of exams and/or the chepest/safest exams.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of arrhythmias in NICMs | At 1 year
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of arrhythmias in NICMs | At 3 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of arrhythmias in NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of arrhythmias in NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of arrhythmias in NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of arrhythmias in NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of arrhythmias in NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of arrhythmias in NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the predictive value of electrophysiological study and electroanatomical arrhythmogenic substrates in risk stratification of NICMs | At 1 year
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the predictive value of electrophysiological study and electroanatomical arrhythmogenic substrates in risk stratification of NICMs | At 3 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the predictive value of electrophysiological study and electroanatomical arrhythmogenic substrates in risk stratification of NICMs | At 5 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the predictive value of electrophysiological study and electroanatomical arrhythmogenic substrates in risk stratification of NICMs | At 10 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the predictive value of electrophysiological study and electroanatomical arrhythmogenic substrates in risk stratification of NICMs | At 15 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the predictive value of electrophysiological study and electroanatomical arrhythmogenic substrates in risk stratification of NICMs | At 20 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the predictive value of electrophysiological study and electroanatomical arrhythmogenic substrates in risk stratification of NICMs | At 25 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the predictive value of electrophysiological study and electroanatomical arrhythmogenic substrates in risk stratification of NICMs | At 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of M-Infl in NICMs, i.e. association with major events | At 1 year
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of M-Infl in NICMs, i.e. association with major events | At 3 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of M-Infl in NICMs, i.e. association with major events | At 5 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of M-Infl in NICMs, i.e. association with major events | At 10 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of M-Infl in NICMs, i.e. association with major events | At 15 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of M-Infl in NICMs, i.e. association with major events | At 20 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of M-Infl in NICMs, i.e. association with major events | At 25 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of the prognostic value of M-Infl in NICMs, i.e. association with major events | At 30 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of the reproducibility of existing risk factors and risk stratification scores for NICMs in a real-world population, i.e. verification of their role in predicting major events | At 1 year
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of the reproducibility of existing risk factors and risk stratification scores for NICMs in a real-world population, i.e. verification of their role in predicting major events | At 3 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of the reproducibility of existing risk factors and risk stratification scores for NICMs in a real-world population, i.e. verification of their role in predicting major events | At 5 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of the reproducibility of existing risk factors and risk stratification scores for NICMs in a real-world population, i.e. verification of their role in predicting major events | At 10 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of the reproducibility of existing risk factors and risk stratification scores for NICMs in a real-world population, i.e. verification of their role in predicting major events | At 15 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of the reproducibility of existing risk factors and risk stratification scores for NICMs in a real-world population, i.e. verification of their role in predicting major events | At 20 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of the reproducibility of existing risk factors and risk stratification scores for NICMs in a real-world population, i.e. verification of their role in predicting major events | At 25 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of the reproducibility of existing risk factors and risk stratification scores for NICMs in a real-world population, i.e. verification of their role in predicting major events | At 30 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Refinement of risk factors and risk stratification scores for NICMs, i.e. working out of models integrating known and new risk factors for the prediction of major events | At 1 year
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Refinement of risk factors and risk stratification scores for NICMs, i.e. working out of models integrating known and new risk factors for the prediction of major events | At 3 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Refinement of risk factors and risk stratification scores for NICMs, i.e. working out of models integrating known and new risk factors for the prediction of major events | At 5 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Refinement of risk factors and risk stratification scores for NICMs, i.e. working out of models integrating known and new risk factors for the prediction of major events | At 10 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Refinement of risk factors and risk stratification scores for NICMs, i.e. working out of models integrating known and new risk factors for the prediction of major events | At 15 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Refinement of risk factors and risk stratification scores for NICMs, i.e. working out of models integrating known and new risk factors for the prediction of major events | At 20 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Refinement of risk factors and risk stratification scores for NICMs, i.e. working out of models integrating known and new risk factors for the prediction of major events | At 25 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Refinement of risk factors and risk stratification scores for NICMs, i.e. working out of models integrating known and new risk factors for the prediction of major events | At 30 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Elaboration of new risk scores for NICMs, also based on modern technologies of machine learning and artificial intelligence, by identifying the most effective combination of prognostic variables capable of predicting major events | At 1 year
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Elaboration of new risk scores for NICMs, also based on modern technologies of machine learning and artificial intelligence, by identifying the most effective combination of prognostic variables capable of predicting major events | At 3 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Elaboration of new risk scores for NICMs, also based on modern technologies of machine learning and artificial intelligence, by identifying the most effective combination of prognostic variables capable of predicting major events | At 5 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Elaboration of new risk scores for NICMs, also based on modern technologies of machine learning and artificial intelligence, by identifying the most effective combination of prognostic variables capable of predicting major events | At 10 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Elaboration of new risk scores for NICMs, also based on modern technologies of machine learning and artificial intelligence, by identifying the most effective combination of prognostic variables capable of predicting major events | At 15 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Elaboration of new risk scores for NICMs, also based on modern technologies of machine learning and artificial intelligence, by identifying the most effective combination of prognostic variables capable of predicting major events | At 20 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Elaboration of new risk scores for NICMs, also based on modern technologies of machine learning and artificial intelligence, by identifying the most effective combination of prognostic variables capable of predicting major events | At 25 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Elaboration of new risk scores for NICMs, also based on modern technologies of machine learning and artificial intelligence, by identifying the most effective combination of prognostic variables capable of predicting major events | At 30 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of new models in control patient cohorts, i.e. verification of their role in predicting major events | At 1 year
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of new models in control patient cohorts, i.e. verification of their role in predicting major events | At 3 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of new models in control patient cohorts, i.e. verification of their role in predicting major events | At 5 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of new models in control patient cohorts, i.e. verification of their role in predicting major events | At 10 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of new models in control patient cohorts, i.e. verification of their role in predicting major events | At 15 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of new models in control patient cohorts, i.e. verification of their role in predicting major events | At 20 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of new models in control patient cohorts, i.e. verification of their role in predicting major events | At 25 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Validation of new models in control patient cohorts, i.e. verification of their role in predicting major events | At 30 years
  Major events include all-cause death, cardiac death, extra-cardiac disease related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Assessment of epidemiology signatures in DCM | At baseline
Assessment of epidemiology signatures in DCM | At 5 years
Assessment of epidemiology signatures in DCM | At 10 years
Assessment of epidemiology signatures in DCM | At 15 years
Assessment of epidemiology signatures in DCM | At 20 years
Assessment of epidemiology signatures in DCM | At 25 years
Assessment of epidemiology signatures in DCM | At 30 years
Assessment of epidemiology signatures in HCM | At baseline
Assessment of epidemiology signatures in HCM | At 5 years
Assessment of epidemiology signatures in HCM | At 10 years
Assessment of epidemiology signatures in HCM | At 15 years
Assessment of epidemiology signatures in HCM | At 20 years
Assessment of epidemiology signatures in HCM | At 25 years
Assessment of epidemiology signatures in HCM | At 30 years
Assessment of epidemiology signatures in RCM | At baseline
Assessment of epidemiology signatures in RCM | At 5 years
Assessment of epidemiology signatures in RCM | At 10 years
Assessment of epidemiology signatures in RCM | At 15 years
Assessment of epidemiology signatures in RCM | At 20 years
Assessment of epidemiology signatures in RCM | At 25 years
Assessment of epidemiology signatures in RCM | At 30 years
Assessment of epidemiology signatures in ACM | At baseline
Assessment of epidemiology signatures in ACM | At 5 years
Assessment of epidemiology signatures in ACM | At 10 years
Assessment of epidemiology signatures in ACM | At 15 years
Assessment of epidemiology signatures in ACM | At 20 years
Assessment of epidemiology signatures in ACM | At 25 years
Assessment of epidemiology signatures in ACM | At 30 years
Assessment of epidemiology signatures in LVNC | At baseline
Assessment of epidemiology signatures in LVNC | At 5 years
Assessment of epidemiology signatures in LVNC | At 10 years
Assessment of epidemiology signatures in LVNC | At 15 years
Assessment of epidemiology signatures in LVNC | At 20 years
Assessment of epidemiology signatures in LVNC | At 25 years
Assessment of epidemiology signatures in LVNC | At 30 years
Assessment of epidemiology signatures in AMVP | At baseline
Assessment of epidemiology signatures in AMVP | At 5 years
Assessment of epidemiology signatures in AMVP | At 10 years
Assessment of epidemiology signatures in AMVP | At 15 years
Assessment of epidemiology signatures in AMVP | At 20 years
Assessment of epidemiology signatures in AMVP | At 25 years
Assessment of epidemiology signatures in AMVP | At 30 years
Assessment of epidemiology signatures in PPCM | At baseline
Assessment of epidemiology signatures in PPCM | At 5 years
Assessment of epidemiology signatures in PPCM | At 10 years
Assessment of epidemiology signatures in PPCM | At 15 years
Assessment of epidemiology signatures in PPCM | At 20 years
Assessment of epidemiology signatures in PPCM | At 25 years
Assessment of epidemiology signatures in PPCM | At 30 years
Assessment of epidemiology signatures in AFD | At baseline
Assessment of epidemiology signatures in AFD | At 5 years
Assessment of epidemiology signatures in AFD | At 10 years
Assessment of epidemiology signatures in AFD | At 15 years
Assessment of epidemiology signatures in AFD | At 20 years
Assessment of epidemiology signatures in AFD | At 25 years
Assessment of epidemiology signatures in AFD | At 30 years
Assessment of epidemiology signatures in storage and dysmetabolic diseases | At baseline
Assessment of epidemiology signatures in storage and dysmetabolic diseases | At 5 years
Assessment of epidemiology signatures in storage and dysmetabolic diseases | At 10 years
Assessment of epidemiology signatures in storage and dysmetabolic diseases | At 15 years
Assessment of epidemiology signatures in storage and dysmetabolic diseases | At 20 years
Assessment of epidemiology signatures in storage and dysmetabolic diseases | At 25 years
Assessment of epidemiology signatures in storage and dysmetabolic diseases | At 30 years
Assessment of epidemiology signatures in mitochondrial diseases | At baseline
Assessment of epidemiology signatures in mitochondrial diseases | At 5 years
Assessment of epidemiology signatures in mitochondrial diseases | At 10 years
Assessment of epidemiology signatures in mitochondrial diseases | At 15 years
Assessment of epidemiology signatures in mitochondrial diseases | At 20 years
Assessment of epidemiology signatures in mitochondrial diseases | At 25 years
Assessment of epidemiology signatures in mitochondrial diseases | At 30 years
Assessment of epidemiology signatures in channelopathies with structural changes | At baseline
Assessment of epidemiology signatures in channelopathies with structural changes | At 5 years
Assessment of epidemiology signatures in channelopathies with structural changes | At 10 years
Assessment of epidemiology signatures in channelopathies with structural changes | At 15 years
Assessment of epidemiology signatures in channelopathies with structural changes | At 20 years
Assessment of epidemiology signatures in channelopathies with structural changes | At 25 years
Assessment of epidemiology signatures in channelopathies with structural changes | At 30 years
Assessment of epidemiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
Assessment of epidemiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
Assessment of epidemiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
Assessment of epidemiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
Assessment of epidemiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
Assessment of epidemiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
Assessment of epidemiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
Assessment of epidemiology signatures in overlapping and undefined phenotypes | At baseline
Assessment of epidemiology signatures in overlapping and undefined phenotypes | At 5 years
Assessment of epidemiology signatures in overlapping and undefined phenotypes | At 10 years
Assessment of epidemiology signatures in overlapping and undefined phenotypes | At 15 years
Assessment of epidemiology signatures in overlapping and undefined phenotypes | At 20 years
Assessment of epidemiology signatures in overlapping and undefined phenotypes | At 25 years
Assessment of epidemiology signatures in overlapping and undefined phenotypes | At 30 years
Assessment of etiology signatures in DCM | At baseline
Assessment of etiology signatures in DCM | At 5 years
Assessment of etiology signatures in DCM | At 10 years
Assessment of etiology signatures in DCM | At 15 years
Assessment of etiology signatures in DCM | At 20 years
Assessment of etiology signatures in DCM | At 25 years
Assessment of etiology signatures in DCM | At 30 years
Assessment of etiology signatures in HCM | At baseline
Assessment of etiology signatures in HCM | At 5 years
Assessment of etiology signatures in HCM | At 10 years
Assessment of etiology signatures in HCM | At 15 years
Assessment of etiology signatures in HCM | At 20 years
Assessment of etiology signatures in HCM | At 25 years
Assessment of etiology signatures in HCM | At 30 years
Assessment of etiology signatures in RCM | At baseline
Assessment of etiology signatures in RCM | At 5 years
Assessment of etiology signatures in RCM | At 10 years
Assessment of etiology signatures in RCM | At 15 years
Assessment of etiology signatures in RCM | At 20 years
Assessment of etiology signatures in RCM | At 25 years
Assessment of etiology signatures in RCM | At 30 years
Assessment of etiology signatures in ACM | At baseline
Assessment of etiology signatures in ACM | At 5 years
Assessment of etiology signatures in ACM | At 10 years
Assessment of etiology signatures in ACM | At 15 years
Assessment of etiology signatures in ACM | At 20 years
Assessment of etiology signatures in ACM | At 25 years
Assessment of etiology signatures in ACM | At 30 years
Assessment of etiology signatures in LVNC | At baseline
Assessment of etiology signatures in LVNC | At 5 years
Assessment of etiology signatures in LVNC | At 10 years
Assessment of etiology signatures in LVNC | At 15 years
Assessment of etiology signatures in LVNC | At 20 years
Assessment of etiology signatures in LVNC | At 25 years
Assessment of etiology signatures in LVNC | At 30 years
Assessment of etiology signatures in AMVP | At baseline
Assessment of etiology signatures in AMVP | At 5 years
Assessment of etiology signatures in AMVP | At 10 years
Assessment of etiology signatures in AMVP | At 15 years
Assessment of etiology signatures in AMVP | At 20 years
Assessment of etiology signatures in AMVP | At 25 years
Assessment of etiology signatures in AMVP | At 30 years
Assessment of etiology signatures in PPCM | At baseline
Assessment of etiology signatures in PPCM | At 5 years
Assessment of etiology signatures in PPCM | At 10 years
Assessment of etiology signatures in PPCM | At 15 years
Assessment of etiology signatures in PPCM | At 20 years
Assessment of etiology signatures in PPCM | At 25 years
Assessment of etiology signatures in PPCM | At 30 years
Assessment of etiology signatures in AFD | At baseline
Assessment of etiology signatures in AFD | At 5 years
Assessment of etiology signatures in AFD | At 10 years
Assessment of etiology signatures in AFD | At 15 years
Assessment of etiology signatures in AFD | At 20 years
Assessment of etiology signatures in AFD | At 25 years
Assessment of etiology signatures in AFD | At 30 years
Assessment of etiology signatures in storage and dysmetabolic diseases | At baseline
Assessment of etiology signatures in storage and dysmetabolic diseases | At 5 years
Assessment of etiology signatures in storage and dysmetabolic diseases | At 10 years
Assessment of etiology signatures in storage and dysmetabolic diseases | At 15 years
Assessment of etiology signatures in storage and dysmetabolic diseases | At 20 years
Assessment of etiology signatures in storage and dysmetabolic diseases | At 25 years
Assessment of etiology signatures in storage and dysmetabolic diseases | At 30 years
Assessment of etiology signatures in mitochondrial diseases | At baseline
Assessment of etiology signatures in mitochondrial diseases | At 5 years
Assessment of etiology signatures in mitochondrial diseases | At 10 years
Assessment of etiology signatures in mitochondrial diseases | At 15 years
Assessment of etiology signatures in mitochondrial diseases | At 20 years
Assessment of etiology signatures in mitochondrial diseases | At 25 years
Assessment of etiology signatures in mitochondrial diseases | At 30 years
Assessment of etiology signatures in channelopathies with structural changes | At baseline
Assessment of etiology signatures in channelopathies with structural changes | At 5 years
Assessment of etiology signatures in channelopathies with structural changes | At 10 years
Assessment of etiology signatures in channelopathies with structural changes | At 15 years
Assessment of etiology signatures in channelopathies with structural changes | At 20 years
Assessment of etiology signatures in channelopathies with structural changes | At 25 years
Assessment of etiology signatures in channelopathies with structural changes | At 30 years
Assessment of etiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
Assessment of etiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
Assessment of etiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
Assessment of etiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
Assessment of etiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
Assessment of etiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
Assessment of etiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
Assessment of etiology signatures in overlapping and undefined phenotypes | At 5 years
Assessment of etiology signatures in overlapping and undefined phenotypes | At 10 years
Assessment of etiology signatures in overlapping and undefined phenotypes | At 15 years
Assessment of etiology signatures in overlapping and undefined phenotypes | At 20 years
Assessment of etiology signatures in overlapping and undefined phenotypes | At 25 years
Assessment of etiology signatures in overlapping and undefined phenotypes | At 30 years
Assessment of pathophysiology signatures in DCM | At baseline
Assessment of pathophysiology signatures in DCM | At 5 years
Assessment of pathophysiology signatures in DCM | At 10 years
Assessment of pathophysiology signatures in DCM | At 15 years
Assessment of pathophysiology signatures in DCM | At 20 years
Assessment of pathophysiology signatures in DCM | At 25 years
Assessment of pathophysiology signatures in DCM | At 30 years
Assessment of pathophysiology signatures in HCM | At baseline
Assessment of pathophysiology signatures in HCM | At 5 years
Assessment of pathophysiology signatures in HCM | At 10 years
Assessment of pathophysiology signatures in HCM | At 15 years
Assessment of pathophysiology signatures in HCM | At 20 years
Assessment of pathophysiology signatures in HCM | At 25 years
Assessment of pathophysiology signatures in HCM | At 30 years
Assessment of pathophysiology signatures in RCM | At baseline
Assessment of pathophysiology signatures in RCM | At 5 years
Assessment of pathophysiology signatures in RCM | At 10 years
Assessment of pathophysiology signatures in RCM | At 15 years
Assessment of pathophysiology signatures in RCM | At 20 years
Assessment of pathophysiology signatures in RCM | At 25 years
Assessment of pathophysiology signatures in RCM | At 30 years
Assessment of pathophysiology signatures in ACM | At baseline
Assessment of pathophysiology signatures in ACM | At 5 years
Assessment of pathophysiology signatures in ACM | At 10 years
Assessment of pathophysiology signatures in ACM | At 15 years
Assessment of pathophysiology signatures in ACM | At 20 years
Assessment of pathophysiology signatures in ACM | At 25 years
Assessment of pathophysiology signatures in ACM | At 30 years
Assessment of pathophysiology signatures in LVNC | At baseline
Assessment of pathophysiology signatures in LVNC | At 5 years
Assessment of pathophysiology signatures in LVNC | At 10 years
Assessment of pathophysiology signatures in LVNC | At 15 years
Assessment of pathophysiology signatures in LVNC | At 20 years
Assessment of pathophysiology signatures in LVNC | At 25 years
Assessment of pathophysiology signatures in LVNC | At 30 years
Assessment of pathophysiology signatures in AMVP | At baseline
Assessment of pathophysiology signatures in AMVP | At 5 years
Assessment of pathophysiology signatures in AMVP | At 10 years
Assessment of pathophysiology signatures in AMVP | At 15 years
Assessment of pathophysiology signatures in AMVP | At 20 years
Assessment of pathophysiology signatures in AMVP | At 25 years
Assessment of pathophysiology signatures in AMVP | At 30 years
Assessment of pathophysiology signatures in PPCM | At baseline
Assessment of pathophysiology signatures in PPCM | At 5 years
Assessment of pathophysiology signatures in PPCM | At 10 years
Assessment of pathophysiology signatures in PPCM | At 15 years
Assessment of pathophysiology signatures in PPCM | At 20 years
Assessment of pathophysiology signatures in PPCM | At 25 years
Assessment of pathophysiology signatures in PPCM | At 30 years
Assessment of pathophysiology signatures in AFD | At baseline
Assessment of pathophysiology signatures in AFD | At 5 years
Assessment of pathophysiology signatures in AFD | At 10 years
Assessment of pathophysiology signatures in AFD | At 15 years
Assessment of pathophysiology signatures in AFD | At 20 years
Assessment of pathophysiology signatures in AFD | At 25 years
Assessment of pathophysiology signatures in AFD | At 30 years
Assessment of pathophysiology signatures in storage and dysmetabolic diseases | At baseline
Assessment of pathophysiology signatures in storage and dysmetabolic diseases | At 5 years
Assessment of pathophysiology signatures in storage and dysmetabolic diseases | At 10 years
Assessment of pathophysiology signatures in storage and dysmetabolic diseases | At 15 years
Assessment of pathophysiology signatures in storage and dysmetabolic diseases | At 20 years
Assessment of pathophysiology signatures in storage and dysmetabolic diseases | At 25 years
Assessment of pathophysiology signatures in storage and dysmetabolic diseases | At 30 years
Assessment of pathophysiology signatures in mitochondrial diseases | At baseline
Assessment of pathophysiology signatures in mitochondrial diseases | At 5 years
Assessment of pathophysiology signatures in mitochondrial diseases | At 10 years
Assessment of pathophysiology signatures in mitochondrial diseases | At 15 years
Assessment of pathophysiology signatures in mitochondrial diseases | At 20 years
Assessment of pathophysiology signatures in mitochondrial diseases | At 25 years
Assessment of pathophysiology signatures in mitochondrial diseases | At 30 years
Assessment of pathophysiology signatures in channelopathies with structural changes | At baseline
Assessment of pathophysiology signatures in channelopathies with structural changes | At 5 years
Assessment of pathophysiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
Assessment of pathophysiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
Assessment of pathophysiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
Assessment of pathophysiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
Assessment of pathophysiology signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
Assessment of pathophysiology signatures in overlapping and undefined phenotypes | At baseline
Assessment of pathophysiology signatures in overlapping and undefined phenotypes | At 5 years
Assessment of pathophysiology signatures in overlapping and undefined phenotypes | At 10 years
Assessment of pathophysiology signatures in overlapping and undefined phenotypes | At 15 years
Assessment of pathophysiology signatures in overlapping and undefined phenotypes | At 20 years
Assessment of pathophysiology signatures in overlapping and undefined phenotypes | At 25 years
Assessment of pathophysiology signatures in overlapping and undefined phenotypes | At 30 years
Assessment of genotype-phenotype signatures in DCM | At baseline
Assessment of genotype-phenotype signatures in DCM | At 5 years
Assessment of genotype-phenotype signatures in DCM | At 10 years
Assessment of genotype-phenotype signatures in DCM | At 15 years
Assessment of genotype-phenotype signatures in DCM | At 20 years
Assessment of genotype-phenotype signatures in DCM | At 25 years
Assessment of genotype-phenotype signatures in DCM | At 30 years
Assessment of genotype-phenotype signatures in HCM | At baseline
Assessment of genotype-phenotype signatures in HCM | At 5 years
Assessment of genotype-phenotype signatures in HCM | At 10 years
Assessment of genotype-phenotype signatures in HCM | At 15 years
Assessment of genotype-phenotype signatures in HCM | At 20 years
Assessment of genotype-phenotype signatures in HCM | At 25 years
Assessment of genotype-phenotype signatures in HCM | At 30 years
Assessment of genotype-phenotype signatures in RCM | At baseline
Assessment of genotype-phenotype signatures in RCM | At 5 years
Assessment of genotype-phenotype signatures in RCM | At 10 years
Assessment of genotype-phenotype signatures in RCM | At 15 years
Assessment of genotype-phenotype signatures in RCM | At 20 years
Assessment of genotype-phenotype signatures in RCM | At 25 years
Assessment of genotype-phenotype signatures in RCM | At 30 years
Assessment of genotype-phenotype signatures in ACM | At baseline
Assessment of genotype-phenotype signatures in ACM | At 5 years
Assessment of genotype-phenotype signatures in ACM | At 10 years
Assessment of genotype-phenotype signatures in ACM | At 15 years
Assessment of genotype-phenotype signatures in ACM | At 20 years
Assessment of genotype-phenotype signatures in ACM | At 25 years
Assessment of genotype-phenotype signatures in ACM | At 30 years
Assessment of genotype-phenotype signatures in LVNC | At baseline
Assessment of genotype-phenotype signatures in LVNC | At 5 years
Assessment of genotype-phenotype signatures in LVNC | At 10 years
Assessment of genotype-phenotype signatures in LVNC | At 15 years
Assessment of genotype-phenotype signatures in LVNC | At 20 years
Assessment of genotype-phenotype signatures in LVNC | At 25 years
Assessment of genotype-phenotype signatures in LVNC | At 30 years
Assessment of genotype-phenotype signatures in AMVP | At baseline
Assessment of genotype-phenotype signatures in AMVP | At 5 years
Assessment of genotype-phenotype signatures in AMVP | At 10 years
Assessment of genotype-phenotype signatures in AMVP | At 15 years
Assessment of genotype-phenotype signatures in AMVP | At 20 years
Assessment of genotype-phenotype signatures in AMVP | At 25 years
Assessment of genotype-phenotype signatures in AMVP | At 30 years
Assessment of genotype-phenotype signatures in PPCM | At baseline
Assessment of genotype-phenotype signatures in PPCM | At 5 years
Assessment of genotype-phenotype signatures in PPCM | At 10 years
Assessment of genotype-phenotype signatures in PPCM | At 15 years
Assessment of genotype-phenotype signatures in PPCM | At 20 years
Assessment of genotype-phenotype signatures in PPCM | At 25 years
Assessment of genotype-phenotype signatures in PPCM | At 30 years
Assessment of genotype-phenotype signatures in AFD | At baseline
Assessment of genotype-phenotype signatures in AFD | At 5 years
Assessment of genotype-phenotype signatures in AFD | At 10 years
Assessment of genotype-phenotype signatures in AFD | At 15 years
Assessment of genotype-phenotype signatures in AFD | At 20 years
Assessment of genotype-phenotype signatures in AFD | At 25 years
Assessment of genotype-phenotype signatures in AFD | At 30 years
Assessment of genotype-phenotype signatures in storage and dysmetabolic diseases | At baseline
Assessment of genotype-phenotype signatures in storage and dysmetabolic diseases | At 5 years
Assessment of genotype-phenotype signatures in storage and dysmetabolic diseases | At 10 years
Assessment of genotype-phenotype signatures in storage and dysmetabolic diseases | At 15 years
Assessment of genotype-phenotype signatures in storage and dysmetabolic diseases | At 20 years
Assessment of genotype-phenotype signatures in storage and dysmetabolic diseases | At 25 years
Assessment of genotype-phenotype signatures in storage and dysmetabolic diseases | At 30 years
Assessment of genotype-phenotype signatures in mitochondrial diseases | At baseline
Assessment of genotype-phenotype signatures in mitochondrial diseases | At 5 years
Assessment of genotype-phenotype signatures in mitochondrial diseases | At 10 years
Assessment of genotype-phenotype signatures in mitochondrial diseases | At 15 years
Assessment of genotype-phenotype signatures in mitochondrial diseases | At 20 years
Assessment of genotype-phenotype signatures in mitochondrial diseases | At 25 years
Assessment of genotype-phenotype signatures in mitochondrial diseases | At 30 years
Assessment of genotype-phenotype signatures in channelopathies with structural changes | At baseline
Assessment of genotype-phenotype signatures in channelopathies with structural changes | At 5 years
Assessment of genotype-phenotype signatures in channelopathies with structural changes | At 10 years
Assessment of genotype-phenotype signatures in channelopathies with structural changes | At 15 years
Assessment of genotype-phenotype signatures in channelopathies with structural changes | At 20 years
Assessment of genotype-phenotype signatures in channelopathies with structural changes | At 25 years
Assessment of genotype-phenotype signatures in channelopathies with structural changes | At 30 years
Assessment of genotype-phenotype signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
Assessment of genotype-phenotype signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
Assessment of genotype-phenotype signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
Assessment of genotype-phenotype signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
Assessment of genotype-phenotype signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
Assessment of genotype-phenotype signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
Assessment of genotype-phenotype signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
Assessment of genotype-phenotype signatures in overlapping and undefined phenotypes | At baseline
Assessment of genotype-phenotype signatures in overlapping and undefined phenotypes | At 5 years
Assessment of genotype-phenotype signatures in overlapping and undefined phenotypes | At 10 years
Assessment of genotype-phenotype signatures in overlapping and undefined phenotypes | At 15 years
Assessment of genotype-phenotype signatures in overlapping and undefined phenotypes | At 20 years
Assessment of genotype-phenotype signatures in overlapping and undefined phenotypes | At 25 years
Assessment of genotype-phenotype signatures in overlapping and undefined phenotypes | At 30 years
Assessment of arrhythmia signatures in DCM | At baseline
Assessment of arrhythmia signatures in DCM | At 5 years
Assessment of arrhythmia signatures in DCM | At 10 years
Assessment of arrhythmia signatures in DCM | At 15 years
Assessment of arrhythmia signatures in DCM | At 20 years
Assessment of arrhythmia signatures in DCM | At 25 years
Assessment of arrhythmia signatures in DCM | At 30 years
Assessment of arrhythmia signatures in HCM | At baseline
Assessment of arrhythmia signatures in HCM | At 5 years
Assessment of arrhythmia signatures in RCM | Every 10 years
Assessment of arrhythmia signatures in ACM | Every 15 years
Assessment of arrhythmia signatures in ACM | Every 20 years
Assessment of arrhythmia signatures in ACM | Every 25 years
Assessment of arrhythmia signatures in ACM | Every 30 years
Assessment of arrhythmia signatures in LVNC | At baseline
Assessment of arrhythmia signatures in LVNC | At 5 years
Assessment of arrhythmia signatures in LVNC | At 10 years
Assessment of arrhythmia signatures in LVNC | At 15 years
Assessment of arrhythmia signatures in LVNC | At 20 years
Assessment of arrhythmia signatures in LVNC | At 25 years
Assessment of arrhythmia signatures in LVNC | At 30 years
Assessment of arrhythmia signatures in AMVP | At baseline
Assessment of arrhythmia signatures in AMVP | At 5 years
Assessment of arrhythmia signatures in AMVP | At 10 years
Assessment of arrhythmia signatures in AMVP | At 15 years
Assessment of arrhythmia signatures in AMVP | At 20 years
Assessment of arrhythmia signatures in AMVP | At 25 years
Assessment of arrhythmia signatures in AMVP | At 30 years
Assessment of arrhythmia signatures in PPCM | At baseline
Assessment of arrhythmia signatures in PPCM | At 5 years
Assessment of arrhythmia signatures in PPCM | At 10 years
Assessment of arrhythmia signatures in PPCM | At 15 years
Assessment of arrhythmia signatures in PPCM | At 20 years
Assessment of arrhythmia signatures in PPCM | At 25 years
Assessment of arrhythmia signatures in PPCM | At 30 years
Assessment of arrhythmia signatures in AFD | At baseline
Assessment of arrhythmia signatures in AFD | At 5 years
Assessment of arrhythmia signatures in AFD | At 10 years
Assessment of arrhythmia signatures in AFD | At 15 years
Assessment of arrhythmia signatures in AFD | At 20 years
Assessment of arrhythmia signatures in AFD | At 25 years
Assessment of arrhythmia signatures in AFD | At 30 years
Assessment of arrhythmia signatures in storage and dysmetabolic diseases | At baseline
Assessment of arrhythmia signatures in storage and dysmetabolic diseases | At 5 years
Assessment of arrhythmia signatures in storage and dysmetabolic diseases | At 10 years
Assessment of arrhythmia signatures in storage and dysmetabolic diseases | At 15 years
Assessment of arrhythmia signatures in storage and dysmetabolic diseases | At 20 years
Assessment of arrhythmia signatures in storage and dysmetabolic diseases | At 25 years
Assessment of arrhythmia signatures in storage and dysmetabolic diseases | At 30 years
Assessment of arrhythmia signatures in mitochondrial diseases | At baseline
Assessment of arrhythmia signatures in mitochondrial diseases | At 5 years
Assessment of arrhythmia signatures in mitochondrial diseases | At 10 years
Assessment of arrhythmia signatures in mitochondrial diseases | At 15 years
Assessment of arrhythmia signatures in mitochondrial diseases | At 20 years
Assessment of arrhythmia signatures in mitochondrial diseases | At 25 years
Assessment of arrhythmia signatures in mitochondrial diseases | At 30 years
Assessment of arrhythmia signatures in channelopathies with structural changes | At baseline
Assessment of arrhythmia signatures in channelopathies with structural changes | At 5 years
Assessment of arrhythmia signatures in channelopathies with structural changes | At 10 years
Assessment of arrhythmia signatures in channelopathies with structural changes | At 15 years
Assessment of arrhythmia signatures in channelopathies with structural changes | At 20 years
Assessment of arrhythmia signatures in channelopathies with structural changes | At 25 years
Assessment of arrhythmia signatures in channelopathies with structural changes | At 30 years
Assessment of arrhythmia signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
Assessment of arrhythmia signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
Assessment of arrhythmia signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
Assessment of arrhythmia signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
Assessment of arrhythmia signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
Assessment of arrhythmia signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
Assessment of arrhythmia signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
Assessment of arrhythmia signatures in overlapping and undefined phenotype | At baseline
Assessment of arrhythmia signatures in overlapping and undefined phenotype | At 5 years
Assessment of arrhythmia signatures in overlapping and undefined phenotype | At 10 years
Assessment of arrhythmia signatures in overlapping and undefined phenotype | At 15 years
Assessment of arrhythmia signatures in overlapping and undefined phenotype | At 20 years
Assessment of arrhythmia signatures in overlapping and undefined phenotype | At 25 years
Assessment of arrhythmia signatures in overlapping and undefined phenotype | At 30 years
Assessment of M-Infl signatures in DCM | At baseline
Assessment of M-Infl signatures in DCM | At 5 years
Assessment of M-Infl signatures in DCM | At 10 years
Assessment of M-Infl signatures in DCM | At 15 years
Assessment of M-Infl signatures in DCM | At 20 years
Assessment of M-Infl signatures in DCM | At 25 years
Assessment of M-Infl signatures in DCM | At 30 years
Assessment of M-Infl signatures in HCM | At baseline
Assessment of M-Infl signatures in HCM | At 5 years
Assessment of M-Infl signatures in HCM | At 10 years
Assessment of M-Infl signatures in HCM | At 15 years
Assessment of M-Infl signatures in HCM | At 20 years
Assessment of M-Infl signatures in HCM | At 25 years
Assessment of M-Infl signatures in HCM | At 30 years
Assessment of M-Infl signatures in RCM | At baseline
Assessment of M-Infl signatures in RCM | At 5 years
Assessment of M-Infl signatures in RCM | At 10 years
Assessment of M-Infl signatures in RCM | At 15 years
Assessment of M-Infl signatures in RCM | At 20 years
Assessment of M-Infl signatures in RCM | At 25 years
Assessment of M-Infl signatures in RCM | At 30 years
Assessment of M-Infl signatures in ACM | At baseline
Assessment of M-Infl signatures in ACM | At 5 years
Assessment of M-Infl signatures in ACM | At 10 years
Assessment of M-Infl signatures in ACM | At 15 years
Assessment of M-Infl signatures in ACM | At 20 years
Assessment of M-Infl signatures in ACM | At 25 years
Assessment of M-Infl signatures in ACM | At 30 years
Assessment of M-Infl signatures in LVNC | At baseline
Assessment of M-Infl signatures in LVNC | At 5 years
Assessment of M-Infl signatures in LVNC | At 10 years
Assessment of M-Infl signatures in LVNC | At 15 years
Assessment of M-Infl signatures in LVNC | At 20 years
Assessment of M-Infl signatures in LVNC | At 25 years
Assessment of M-Infl signatures in LVNC | At 30 years
Assessment of M-Infl signatures in AMVP | At baseline
Assessment of M-Infl signatures in AMVP | At 5 years
Assessment of M-Infl signatures in AMVP | At 10 years
Assessment of M-Infl signatures in AMVP | At 15 years
Assessment of M-Infl signatures in AMVP | At 20 years
Assessment of M-Infl signatures in AMVP | At 25 years
Assessment of M-Infl signatures in AMVP | At 30 years
Assessment of M-Infl signatures in PPCM | At baseline
Assessment of M-Infl signatures in PPCM | At 5 years
Assessment of M-Infl signatures in PPCM | At 10 years
Assessment of M-Infl signatures in PPCM | At 15 years
Assessment of M-Infl signatures in PPCM | At 20 years
Assessment of M-Infl signatures in PPCM | At 25 years
Assessment of M-Infl signatures in PPCM | At 30 years
Assessment of M-Infl signatures in AFD | At baseline
Assessment of M-Infl signatures in AFD | At 5 years
Assessment of M-Infl signatures in AFD | At 10 years
Assessment of M-Infl signatures in AFD | At 15 years
Assessment of M-Infl signatures in AFD | At 20 years
Assessment of M-Infl signatures in AFD | At 25 years
Assessment of M-Infl signatures in AFD | At 30 years
Assessment of M-Infl signatures in storage and dysmetabolic diseases | At baseline
Assessment of M-Infl signatures in storage and dysmetabolic diseases | At 5 years
Assessment of M-Infl signatures in storage and dysmetabolic diseases | At 10 years
Assessment of M-Infl signatures in storage and dysmetabolic diseases | At 15 years
Assessment of M-Infl signatures in storage and dysmetabolic diseases | At 20 years
Assessment of M-Infl signatures in storage and dysmetabolic diseases | At 25 years
Assessment of M-Infl signatures in storage and dysmetabolic diseases | At 30 years
Assessment of M-Infl signatures in mitochondrial diseases | At baseline
Assessment of M-Infl signatures in mitochondrial diseases | At 5 years
Assessment of M-Infl signatures in mitochondrial diseases | At 10 years
Assessment of M-Infl signatures in mitochondrial diseases | At 15 years
Assessment of M-Infl signatures in mitochondrial diseases | At 20 years
Assessment of M-Infl signatures in mitochondrial diseases | At 25 years
Assessment of M-Infl signatures in mitochondrial diseases | At 30 years
Assessment of M-Infl signatures in channelopathies with structural changes | At baseline
Assessment of M-Infl signatures in channelopathies with structural changes | At 5 years
Assessment of M-Infl signatures in channelopathies with structural changes | At 10 years
Assessment of M-Infl signatures in channelopathies with structural changes | At 15 years
Assessment of M-Infl signatures in channelopathies with structural changes | At 20 years
Assessment of M-Infl signatures in channelopathies with structural changes | At 25 years
Assessment of M-Infl signatures in channelopathies with structural changes | At 30 years
Assessment of M-Infl signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
Assessment of M-Infl signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
Assessment of M-Infl signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
Assessment of M-Infl signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
Assessment of M-Infl signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
Assessment of M-Infl signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
Assessment of M-Infl signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
Assessment of M-Infl signatures in overlapping and undefined phenotypes | At baseline
Assessment of M-Infl signatures in overlapping and undefined phenotypes | At 5 years
Assessment of M-Infl signatures in overlapping and undefined phenotypes | At 10 years
Assessment of M-Infl signatures in overlapping and undefined phenotypes | At 15 years
Assessment of M-Infl signatures in overlapping and undefined phenotypes | At 20 years
Assessment of M-Infl signatures in overlapping and undefined phenotypes | At 25 years
Assessment of M-Infl signatures in overlapping and undefined phenotypes | At 30 years
Assessment of extracardiac signatures in DCM | At baseline
Assessment of extracardiac signatures in DCM | At 5 years
Assessment of extracardiac signatures in DCM | At 10 years
Assessment of extracardiac signatures in DCM | At 15 years
Assessment of extracardiac signatures in DCM | At 20 years
Assessment of extracardiac signatures in DCM | At 25 years
Assessment of extracardiac signatures in DCM | At 30 years
Assessment of extracardiac signatures in HCM | At baseline
Assessment of extracardiac signatures in HCM | At 5 years
Assessment of extracardiac signatures in HCM | At 10 years
Assessment of extracardiac signatures in HCM | At 15 years
Assessment of extracardiac signatures in HCM | At 20 years
Assessment of extracardiac signatures in HCM | At 25 years
Assessment of extracardiac signatures in HCM | At 30 years
Assessment of extracardiac signatures in RCM | At baseline
Assessment of extracardiac signatures in RCM | At 5 years
Assessment of extracardiac signatures in RCM | At 10 years
Assessment of extracardiac signatures in RCM | At 15 years
Assessment of extracardiac signatures in RCM | At 20 years
Assessment of extracardiac signatures in RCM | At 25 years
Assessment of extracardiac signatures in RCM | At 30 years
Assessment of extracardiac signatures in ACM | At baseline
Assessment of extracardiac signatures in ACM | At 5 years
Assessment of extracardiac signatures in ACM | At 10 years
Assessment of extracardiac signatures in ACM | At 15 years
Assessment of extracardiac signatures in ACM | At 20 years
Assessment of extracardiac signatures in ACM | At 25 years
Assessment of extracardiac signatures in ACM | At 30 years
Assessment of extracardiac signatures in LVNC | At baseline
Assessment of extracardiac signatures in LVNC | At 5 years
Assessment of extracardiac signatures in LVNC | At 10 years
Assessment of extracardiac signatures in LVNC | At 15 years
Assessment of extracardiac signatures in LVNC | At 20 years
Assessment of extracardiac signatures in LVNC | At 25 years
Assessment of extracardiac signatures in LVNC | At 30 years
Assessment of extracardiac signatures in AMVP | At baseline
Assessment of extracardiac signatures in AMVP | At 5 years
Assessment of extracardiac signatures in AMVP | At 10 years
Assessment of extracardiac signatures in AMVP | At 15 years
Assessment of extracardiac signatures in AMVP | At 20 years
Assessment of extracardiac signatures in AMVP | At 25 years
Assessment of extracardiac signatures in AMVP | At 30 years
Assessment of extracardiac signatures in PPCM | At baseline
Assessment of extracardiac signatures in PPCM | At 5 years
Assessment of extracardiac signatures in PPCM | At 10 years
Assessment of extracardiac signatures in PPCM | At 15 years
Assessment of extracardiac signatures in PPCM | At 20 years
Assessment of extracardiac signatures in PPCM | At 25 years
Assessment of extracardiac signatures in PPCM | At 30 years
Assessment of extracardiac signatures in AFD | At baseline
Assessment of extracardiac signatures in AFD | At 5 years
Assessment of extracardiac signatures in AFD | At 10 years
Assessment of extracardiac signatures in AFD | At 15 years
Assessment of extracardiac signatures in AFD | At 20 years
Assessment of extracardiac signatures in AFD | At 25 years
Assessment of extracardiac signatures in AFD | At 30 years
Assessment of extracardiac signatures in storage and dysmetabolic diseases | At baseline
Assessment of extracardiac signatures in storage and dysmetabolic diseases | At 5 years
Assessment of extracardiac signatures in storage and dysmetabolic diseases | At 10 years
Assessment of extracardiac signatures in storage and dysmetabolic diseases | At 15 years
Assessment of extracardiac signatures in storage and dysmetabolic diseases | At 20 years
Assessment of extracardiac signatures in storage and dysmetabolic diseases | At 25 years
Assessment of extracardiac signatures in storage and dysmetabolic diseases | At 30 years
Assessment of extracardiac signatures in mitochondrial diseases | At baseline
Assessment of extracardiac signatures in mitochondrial diseases | At 5 years
Assessment of extracardiac signatures in mitochondrial diseases | At 10 years
Assessment of extracardiac signatures in mitochondrial diseases | At 15 years
Assessment of extracardiac signatures in mitochondrial diseases | At 20 years
Assessment of extracardiac signatures in mitochondrial diseases | At 25 years
Assessment of extracardiac signatures in mitochondrial diseases | At 30 years
Assessment of extracardiac signatures in channelopathies with structural changes | At baseline
Assessment of extracardiac signatures in channelopathies with structural changes | At 5 years
Assessment of extracardiac signatures in channelopathies with structural changes | At 10 years
Assessment of extracardiac signatures in channelopathies with structural changes | At 15 years
Assessment of extracardiac signatures in channelopathies with structural changes | At 20 years
Assessment of extracardiac signatures in channelopathies with structural changes | At 25 years
Assessment of extracardiac signatures in channelopathies with structural changes | At 30 years
Assessment of extracardiac signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
Assessment of extracardiac signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
Assessment of extracardiac signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
Assessment of extracardiac signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
Assessment of extracardiac signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
Assessment of extracardiac signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
Assessment of extracardiac signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
Assessment of extracardiac signatures in overlapping and undefined phenotypes | At baseline
Assessment of extracardiac signatures in overlapping and undefined phenotypes | At 5 years
Assessment of extracardiac signatures in overlapping and undefined phenotypes | At 10 years
Assessment of extracardiac signatures in overlapping and undefined phenotypes | At 15 years
Assessment of extracardiac signatures in overlapping and undefined phenotypes | At 20 years
Assessment of extracardiac signatures in overlapping and undefined phenotypes | At 25 years
Assessment of extracardiac signatures in overlapping and undefined phenotypes | At 30 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in DCM | At baseline
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in DCM | At 5 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in DCM | At 10 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in DCM | At 15 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in DCM | At 20 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in DCM | At 25 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in DCM | At 30 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in HCM | At baseline
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in HCM | At 5 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in HCM | At 10 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in HCM | At 15 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in HCM | At 20 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in HCM | At 25 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in HCM | At 30 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in RCM | At baseline
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in RCM | At 5 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in RCM | At 10 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in RCM | At 15 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in RCM | At 20 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in RCM | At 25 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in RCM | At 30 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in ACM | At baseline
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in ACM | At 5 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in ACM | At 10 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in ACM | At 15 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in ACM | At 20 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in ACM | At 25 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in ACM | At 30 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At baseline
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 5 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 10 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 15 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 20 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 25 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 30 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in overlapping and undefined phenotypes | At baseline
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in overlapping and undefined phenotypes | At 5 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in overlapping and undefined phenotypes | At 10 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in overlapping and undefined phenotypes | At 15 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in overlapping and undefined phenotypes | At 20 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in overlapping and undefined phenotypes | At 25 years
Assessment of multidisciplinary, multimodal, multiparametric diagnostic signatures in overlapping and undefined phenotypes | At 30 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in DCM | At baseline
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in DCM | At 5 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in DCM | At 10 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in DCM | At 15 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in DCM | At 20 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in DCM | At 25 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in DCM | At 30 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in HCM | At baseline
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in HCM | At 5 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in HCM | At 10 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in HCM | At 15 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in HCM | At 20 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in HCM | At 25 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in HCM | At 30 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in RCM | At baseline
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in RCM | At 5 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in RCM | At 10 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in RCM | At 15 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in RCM | At 20 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in RCM | At 25 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in RCM | At 30 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in ACM | At baseline
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in ACM | At 5 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in ACM | At 10 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in ACM | At 15 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in ACM | At 20 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in ACM | At 25 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in ACM | At 30 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in LVNC | At baseline
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in LVNC | At 5 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in LVNC | At 10 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in LVNC | At 15 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in LVNC | At 20 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in LVNC | At 25 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in LVNC | At 30 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AMVP | At baseline
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AMVP | At 5 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AMVP | At 10 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AMVP | At 15 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AMVP | At 20 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AMVP | At 25 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AMVP | At 30 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in PPCM | At baseline
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in PPCM | At 5 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in PPCM | At 10 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in PPCM | At 15 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in PPCM | At 20 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in PPCM | At 25 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in PPCM | At 30 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AFD | At baseline
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AFD | At 5 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AFD | At 10 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AFD | At 15 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AFD | At 20 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AFD | At 25 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in AFD | At 30 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At baseline
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 5 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 10 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 15 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 20 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 25 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | At 30 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in overlapping and undefined phenotypes | At baseline
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in overlapping and undefined phenotypes | At 5 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in overlapping and undefined phenotypes | At 10 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in overlapping and undefined phenotypes | At 15 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in overlapping and undefined phenotypes | At 20 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in overlapping and undefined phenotypes | At 25 years
Assessment of laboratory, tissue, cell, metabolic or multiomic signatures in overlapping and undefined phenotypes | At 30 years
Assessment of prognostic signatures in DCM | At baseline
Assessment of prognostic signatures in DCM | At 5 years
Assessment of prognostic signatures in DCM | At 10 years
Assessment of prognostic signatures in DCM | At 15 years
Assessment of prognostic signatures in DCM | At 20 years
Assessment of prognostic signatures in DCM | At 25 years
Assessment of prognostic signatures in DCM | At 30 years
Assessment of prognostic signatures in HCM | At baseline
Assessment of prognostic signatures in HCM | At 5 years
Assessment of prognostic signatures in HCM | At 10 years
Assessment of prognostic signatures in HCM | At 15 years
Assessment of prognostic signatures in HCM | At 20 years
Assessment of prognostic signatures in HCM | At 25 years
Assessment of prognostic signatures in HCM | At 30 years
Assessment of prognostic signatures in RCM | At baseline
Assessment of prognostic signatures in RCM | At 5 years
Assessment of prognostic signatures in RCM | At 10 years
Assessment of prognostic signatures in RCM | At 15 years
Assessment of prognostic signatures in RCM | At 20 years
Assessment of prognostic signatures in RCM | At 25 years
Assessment of prognostic signatures in RCM | At 30 years
Assessment of prognostic signatures in ACM | At baseline
Assessment of prognostic signatures in ACM | At 5 years
Assessment of prognostic signatures in ACM | At 10 years
Assessment of prognostic signatures in ACM | At 15 years
Assessment of prognostic signatures in ACM | At 20 years
Assessment of prognostic signatures in ACM | At 25 years
Assessment of prognostic signatures in ACM | At 30 years
Assessment of prognostic signatures in LVNC | At baseline
Assessment of prognostic signatures in LVNC | At 5 years
Assessment of prognostic signatures in LVNC | At 10 years
Assessment of prognostic signatures in LVNC | At 15 years
Assessment of prognostic signatures in LVNC | At 20 years
Assessment of prognostic signatures in LVNC | At 25 years
Assessment of prognostic signatures in LVNC | At 30 years
Assessment of prognostic signatures in AMVP | At baseline
Assessment of prognostic signatures in AMVP | At 5 years
Assessment of prognostic signatures in AMVP | At 10 years
Assessment of prognostic signatures in AMVP | At 15 years
Assessment of prognostic signatures in AMVP | At 20 years
Assessment of prognostic signatures in AMVP | At 25 years
Assessment of prognostic signatures in AMVP | At 30 years
Assessment of prognostic signatures in PPCM | At baseline
Assessment of prognostic signatures in PPCM | At 5 years
Assessment of prognostic signatures in PPCM | At 10 years
Assessment of prognostic signatures in PPCM | At 15 years
Assessment of prognostic signatures in PPCM | At 20 years
Assessment of prognostic signatures in PPCM | At 25 years
Assessment of prognostic signatures in PPCM | At 30 years
Assessment of prognostic signatures in AFD | At baseline
Assessment of prognostic signatures in AFD | At 5 years
Assessment of prognostic signatures in AFD | At 10 years
Assessment of prognostic signatures in AFD | At 15 years
Assessment of prognostic signatures in AFD | At 20 years
Assessment of prognostic signatures in AFD | At 25 years
Assessment of prognostic signatures in AFD | At 30 years
Assessment of prognostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
Assessment of prognostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
Assessment of prognostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
Assessment of prognostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
Assessment of prognostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
Assessment of prognostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
Assessment of prognostic signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
Assessment of prognostic signatures in overlapping and undefined phenotypes | At baseline
Assessment of prognostic signatures in overlapping and undefined phenotypes | At 5 years
Assessment of prognostic signatures in overlapping and undefined phenotypes | At 10 years
Assessment of prognostic signatures in overlapping and undefined phenotypes | At 15 years
Assessment of prognostic signatures in overlapping and undefined phenotypes | At 20 years
Assessment of prognostic signatures in overlapping and undefined phenotypes | At 25 years
Assessment of prognostic signatures in overlapping and undefined phenotypes | At 30 years
Assessment of response to treatment signatures in DCM | At baseline
Assessment of response to treatment signatures in DCM | At 5 years
Assessment of response to treatment signatures in DCM | At 10 years
Assessment of response to treatment signatures in DCM | At 15 years
Assessment of response to treatment signatures in DCM | At 20 years
Assessment of response to treatment signatures in DCM | At 25 years
Assessment of response to treatment signatures in DCM | At 30 years
Assessment of response to treatment signatures in HCM | At baseline
Assessment of response to treatment signatures in HCM | At 5 years
Assessment of response to treatment signatures in HCM | At 10 years
Assessment of response to treatment signatures in HCM | At 15 years
Assessment of response to treatment signatures in HCM | At 20 years
Assessment of response to treatment signatures in HCM | At 25 years
Assessment of response to treatment signatures in HCM | At 30 years
Assessment of response to treatment signatures in RCM | At baseline
Assessment of response to treatment signatures in RCM | At 5 years
Assessment of response to treatment signatures in RCM | At 10 years
Assessment of response to treatment signatures in RCM | At 15 years
Assessment of response to treatment signatures in RCM | At 20 years
Assessment of response to treatment signatures in RCM | At 25 years
Assessment of response to treatment signatures in RCM | At 30 years
Assessment of response to treatment signatures in ACM | At baseline
Assessment of response to treatment signatures in ACM | At 5 years
Assessment of response to treatment signatures in ACM | At 10 years
Assessment of response to treatment signatures in ACM | At 15 years
Assessment of response to treatment signatures in ACM | At 20 years
Assessment of response to treatment signatures in ACM | At 25 years
Assessment of response to treatment signatures in ACM | At 30 years
Assessment of response to treatment signatures in LVNC | At baseline
Assessment of response to treatment signatures in LVNC | At 5 years
Assessment of response to treatment signatures in LVNC | At 10 years
Assessment of response to treatment signatures in LVNC | At 15 years
Assessment of response to treatment signatures in LVNC | At 20 years
Assessment of response to treatment signatures in LVNC | At 25 years
Assessment of response to treatment signatures in LVNC | At 30 years
Assessment of response to treatment signatures in AMVP | At baseline
Assessment of response to treatment signatures in AMVP | At 5 years
Assessment of response to treatment signatures in AMVP | At 10 years
Assessment of response to treatment signatures in AMVP | At 15 years
Assessment of response to treatment signatures in AMVP | At 20 years
Assessment of response to treatment signatures in AMVP | At 25 years
Assessment of response to treatment signatures in AMVP | At 30 years
Assessment of response to treatment signatures in PPCM | At baseline
Assessment of response to treatment signatures in PPCM | At 5 years
Assessment of response to treatment signatures in PPCM | At 10 years
Assessment of response to treatment signatures in PPCM | At 15 years
Assessment of response to treatment signatures in PPCM | At 20 years
Assessment of response to treatment signatures in PPCM | At 25 years
Assessment of response to treatment signatures in PPCM | At 30 years
Assessment of response to treatment signatures in AFD | At baseline
Assessment of response to treatment signatures in AFD | At 5 years
Assessment of response to treatment signatures in AFD | At 10 years
Assessment of response to treatment signatures in AFD | At 15 years
Assessment of response to treatment signatures in AFD | At 20 years
Assessment of response to treatment signatures in AFD | At 25 years
Assessment of response to treatment signatures in AFD | At 30 years
Assessment of response to treatment signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
Assessment of response to treatment signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
Assessment of response to treatment signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
Assessment of response to treatment signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
Assessment of response to treatment signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
Assessment of response to treatment signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
Assessment of response to treatment signatures in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes, and cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
Assessment of response to treatment signatures in overlapping and undefined phenotypes | At baseline
Assessment of response to treatment signatures in overlapping and undefined phenotypes | At 5 years
Assessment of response to treatment signatures in overlapping and undefined phenotypes | At 10 years
Assessment of response to treatment signatures in overlapping and undefined phenotypes | At 15 years
Assessment of response to treatment signatures in overlapping and undefined phenotypes | At 20 years
Assessment of response to treatment signatures in overlapping and undefined phenotypes | At 25 years
Assessment of response to treatment signatures in overlapping and undefined phenotypes | At 30 years
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in DCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in DCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in DCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in DCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in DCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in DCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in DCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in HCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in HCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in HCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in HCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in HCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in HCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in HCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in RCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in RCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in RCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in RCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in RCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in RCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in RCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in ACM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in ACM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in ACM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in ACM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in ACM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in ACM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in ACM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in LVNC Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in LVNC Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in LVNC Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in LVNC Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in LVNC Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in LVNC Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in LVNC Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AMVP Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AMVP Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AMVP Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AMVP Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AMVP Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AMVP Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AMVP Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in PPCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in PPCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in PPCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in PPCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in PPCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in PPCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in PPCM Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AFD Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AFD Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AFD Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AFD Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AFD Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AFD Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in AFD Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in storage and dysmetabolic diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in storage and dysmetabolic diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in storage and dysmetabolic diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in storage and dysmetabolic diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in storage and dysmetabolic diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in storage and dysmetabolic diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in storage and dysmetabolic diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in mitochondrial diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in mitochondrial diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in mitochondrial diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in mitochondrial diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in mitochondrial diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in mitochondrial diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in mitochondrial diseases Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in channelopathies with structural changes Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in channelopathies with structural changes Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in channelopathies with structural changes Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in channelopathies with structural changes Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in channelopathies with structural changes Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in channelopathies with structural changes Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in channelopathies with structural changes Efficacy of pharmacological antiarrhythmic treatment on major and minor events | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At baseline
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 5 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 10 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 15 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 20 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 25 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | At 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of pharmacological antiarrhythmic treatment on major and minor events in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Evaluation of efficacy of treatment, defined based on the incidence of minor events during follow-up in overlapping and undefined phenotypes Efficacy of pharmacological antiarrhythmic treatment on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatment on arrhythmic and inflammatory outcomes, as well as on major and minor events in DCM | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatment on arrhythmic and inflammatory outcomes, as well as on major and minor events in HCM | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatment on arrhythmic and inflammatory outcomes, as well as on major and minor events in RCM | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatment on arrhythmic and inflammatory outcomes, as well as on major and minor events in ACM | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatment on arrhythmic and inflammatory outcomes, as well as on major and minor events in LVNC | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatment on arrhythmic and inflammatory outcomes, as well as on major and minor events in AMVP | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatment on arrhythmic and inflammatory outcomes, as well as on major and minor events in PPCM | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatment on arrhythmic and inflammatory outcomes, as well as on major and minor events in AFD | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatment on arrhythmic and inflammatory outcomes, as well as on major and minor events in storage and dysmetabolic diseases, mitochondrial diseases, channelopathies with structural changes | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatment on arrhythmic and inflammatory outcomes, as well as on major and minor events in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatment on arrhythmic and inflammatory outcomes, as well as on major and minor events in overlapping and undefined phenotypes | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Identification of criteria for device implants (PM, ICD, S-ICD, CRT-D...) in NICMs patients | By 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of the most suitable therapeutic strategies based on indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes | By 30 years
  This applies to NICM patients with supraventricular arrhythmias, bradyarrhythmias, or ventricular arrhythmias, with or without M-Inf.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Identification of the best candidates to multidisciplinary management of NICMs | By 30 years
  by identification of the subgroups of patients showing the maximal effects (i.e. lowest incidence of major and minor adverse events) and the minimal risks (i.e. lowest incidence of side effects) following application of multidisciplinary care.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Indication and timing for device (ICD, CRT-D) implant in primary prevention, based on multidisciplinary, multimodal, multiparametric risk assessment in NICMs, and in relation to different general and etiology-dependent treatments | By 30 years
  by identification of the subgroups of patients showing the maximal effects (i.e. lowest incidence of major and minor adverse events) and the minimal risks (i.e. lowest incidence of side effects) following application of multidisciplinary care.
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in DCM patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in HCM patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in RCM patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in ACM patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in LVNC patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in PPCM patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in AMVP patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in AFD patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in storage and dysmetabolic diseases patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in mitochondrial diseases patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in channelopathies with structural changes patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of multidisciplinary patient - tailored approach for the management of inflammation and comorbidities in cardiomyopathies associated with overlapping and undefined phenotypes patients, i.e. effects on major and minor events | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in DCM patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in HCM patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in RCM patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in ACM patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in LVNC patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in AMVP patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in PPCM patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in AFD patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in storage and dysmetabolic diseases patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in mitochondrial diseases patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in channelopathies with structural change patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases patients, , i.e. effects on major and minor events | By 30 years
  Analysis of safety, i.e. incidence of adverse reactions.
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of support treatment, optimal cardiological treatment, and treatment options for heart failure in overlapping and undefined phenotypes patients, , i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in DCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in HCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in RCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in ACM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in LVNC i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in AMVP i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in PPCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in AFD i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in mitochondrial diseases i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in storage and dysmetabolic diseases i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in channelopathies with structural changes i.e. effects on major and minor events. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes).
  Analysis of safety, i.e. incidence of adverse reactions.
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases i.e. effects on major and minor events. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes).
  Analysis of safety, i.e. incidence of adverse reactions.
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of immunomodulatory, immunosuppressive and anti-inflammatory therapy, including biological targeted therapy in overlapping and undefined phenotypes i.e. effects on major and minor events. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes).
  Analysis of safety, i.e. incidence of adverse reactions.
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology -specific treatments, including those aimed to target extra - cardiac disease manifestations in DCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in HCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in RCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in ACM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in LVNC i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in AMVP i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in PPCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in AFD i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in storage and dysmetabolic diseases i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in mitochondrial diseases i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in channelopathies with structural changes i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases i.e. effects on major and minor events. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes) Analysis of safety, i.e. incidence of adverse reactions.
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of etiology-specific treatments, including those aimed to target extra-cardiac disease manifestations in overlapping and undefined phenotypes i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in DCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in HCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in RCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in ACM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in LVNC i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in AMVP i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in PPCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in AFD i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in storage and dysmetabolic diseases, mitochondrial diseases i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in channelopathies with structural changes i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of replacement therapy, molecular therapy, gene therapy in overlapping and undefined phenotypes i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in DCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in HCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in RCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in ACM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in LVNC i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in AMVP i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in PPCM i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in AFD i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in storage and dysmetabolic diseases, mitochondrial diseases i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in channelopathies with structural changes i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases i.e. effects on major and minor events. | By 30 years
  Analysis of safety, i.e. incidence of adverse reactions.
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of heart transplantation and other treatment for end-stage heart failure in overlapping and undefined phenotypes i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in DCM, i.e. effects on major and minor event i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in HCM, i.e. effects on major and minor event i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in RCM, i.e. effects on major and minor event i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in ACM, i.e. effects on major and minor event i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in LVNC, i.e. effects on major and minor event i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in AMVP, i.e. effects on major and minor event i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in PPCM, i.e. effects on major and minor event i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in AFD, i.e. effects on major and minor event i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in storage and dysmetabolic diseases, mitochondrial diseases, i.e. effects on major and minor event i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in channelopathies with structural changes, i.e. effects on major and minor event i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in cardiomyopathies associated with systemic rheumatologic or neuromuscular diseases, i.e. effects on major and minor event i.e. effects on major and minor events. | By 30 years
  Analysis of safety, i.e. incidence of adverse reactions.
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Efficacy of surgical or hemodynamic procedures in overlapping and undefined phenotypes, i.e. effects on major and minor event i.e. effects on major and minor events. Analysis of safety, i.e. incidence of adverse reactions. | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Investigation of cardiac device implant in primary and secondary prevention, in all patients, as well as in subgroups with and without M-Infl in NICMs | By 30 years
  (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes)
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Investigation of ablation of cardiac arrhythmias (indications, patient selection, timing, risk-to-benefit ratio, side effects, duration, challenges, relationships with outcomes) in NICMs | By 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Role of ablation (any technique) on arrhythmic outcomes in NICMs, in all patients, as well as in subgroups with and without arrhythmias and MInfl | By 30 years
  NICMs will include but not limit to: DCM, HCM, RCM, ACM, inflammatory, infiltrative, toxic, dysmetabolic, mitochondrial, neuromuscular, rheumatologic/autoimmune cardiomyopathies, channelopathies with structural substrates, LVNC, PPCM, AMVP, AFD, athlete's heart, undefined and overlap cardiomyopathies. Additional diseases of the NICM spectrum will be included in parallel with the advance of the current knowledge.
Indications and optimal timing for any electrophysiological or interventional procedures in HCM, i.e. comparison of incidence of major and minor events in patients undergoing treatment at different timings | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Indications and optimal timing for any electrophysiological or interventional procedures in ACM, i.e. comparison of incidence of major and minor events in patients undergoing treatment at different timings | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Indications and optimal timing for any electrophysiological or interventional procedures in LVNC, i.e. comparison of incidence of major and minor events in patients undergoing treatment at different timings | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Indications and optimal timing for any electrophysiological or interventional procedures in AMVP, i.e. comparison of incidence of major and minor events in patients undergoing treatment at different timings | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Indications and optimal timing for any electrophysiological or interventional procedures in PPCM, i.e. comparison of incidence of major and minor events in patients undergoing treatment at different timings | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Indications and optimal timing for any electrophysiological or interventional procedures in AFD, i.e. comparison of incidence of major and minor events in patients undergoing treatment at different timings | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Indications and optimal timing for any electrophysiological or interventional procedures in storage and dysmetabolic diseases, i.e. comparison of incidence of major and minor events in patients undergoing treatment at different timings | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Indications and optimal timing for any electrophysiological or interventional procedures in mitochondrial diseases, i.e. comparison of incidence of major and minor events in patients undergoing treatment at different timings | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Indications and optimal timing for any electrophysiological or interventional procedures in channelopathies with structural changes, i.e. comparison of incidence of major and minor events in patients undergoing treatment at different timings | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Indications and optimal timing for any electrophysiological or interventional procedures rheumatologic or neuromuscular diseases | By 30 years
  i.e. comparison of incidence of major and minor events in patients undergoing treatment at different timings.
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.
Indications and optimal timing for any electrophysiological or interventional procedures in overlapping and undefined phenotypes, i.e. comparison of incidence of major and minor events in patients undergoing treatment at different timings | By 30 years
  Major events: all-cause death, cardiac death, extra-cardiac disease-related death, major ventricular arrhythmias (ventricular tachycardia, fibrillation, appropriate ICD therapy), advanced atrioventricular blocks, heart transplantation, end-stage heart failure, disease-related hospitalizations, left/right ventricular systolic dysfunction, presence/persistence/clearance/recurrence of M-Infl.
  Minor events: non-sustained ventricular arrhythmias, supraventricular arrhythmias, other bradyarrhythmias, any structural/functional myocardial abnormality detectable by multimodal diagnostic workup, abnormal laboratory, tissue or multiomic biomarkers, all-cause hospitalizations, disease costs, complications related to disease management, extra-cardiac disease-related non-fatal endpoints.

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Della Bella, MD, Study Chair — San Raffaele Scientific Institute, Milan, Italy
Locations (1):
- IRCCS San Raffaele Scientific Institute, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Requests will be evaluated case by case by the PI.

REFERENCES:
- [Background] Bariani R, Cipriani A, Rizzo S, Celeghin R, Bueno Marinas M, Giorgi B, De Gaspari M, Rigato I, Leoni L, Zorzi A, De Lazzari M, Rampazzo A, Iliceto S, Thiene G, Corrado D, Pilichou K, Basso C, Perazzolo Marra M, Bauce B. 'Hot phase' clinical presentation in arrhythmogenic cardiomyopathy. Europace. 2021 Jun 7;23(6):907-917. doi: 10.1093/europace/euaa343. PMID 33313835
- [Background] Basso C, Thiene G, Corrado D, Angelini A, Nava A, Valente M. Arrhythmogenic right ventricular cardiomyopathy. Dysplasia, dystrophy, or myocarditis? Circulation. 1996 Sep 1;94(5):983-91. doi: 10.1161/01.cir.94.5.983. PMID 8790036
- [Background] Peretto G, De Luca G, Campochiaro C, Palmisano A, Busnardo E, Sartorelli S, Barzaghi F, Cicalese MP, Esposito A, Sala S. Telemedicine in myocarditis: Evolution of a mutidisciplinary "disease unit" at the time of COVID-19 pandemic. Am Heart J. 2020 Nov;229:121-126. doi: 10.1016/j.ahj.2020.07.015. Epub 2020 Aug 12. PMID 32957030
- [Background] Peretto G, Sala S, Della Bella P. [Diagnostic and therapeutic approach to myocarditis patients presenting with arrhythmias]. G Ital Cardiol (Rome). 2020 Mar;21(3):187-194. doi: 10.1714/3306.32767. Italian. PMID 32100731
- [Background] Della Bella P, Baratto F, Vergara P, Bertocchi P, Santamaria M, Notarstefano P, Calo L, Orsida D, Tomasi L, Piacenti M, Sangiorgio S, Pentimalli F, Pruvot E, De Sousa J, Sacher F, Tritto M, Rebellato L, Deneke T, Romano SA, Nesti M, Gargaro A, Giacopelli D, Peretto G, Radinovic A. Does Timing of Ventricular Tachycardia Ablation Affect Prognosis in Patients With an Implantable Cardioverter Defibrillator? Results From the Multicenter Randomized PARTITA Trial. Circulation. 2022 Jun 21;145(25):1829-1838. doi: 10.1161/CIRCULATIONAHA.122.059598. Epub 2022 Apr 3. PMID 35369700
- [Background] Della Bella P, Baratto F, Tsiachris D, Trevisi N, Vergara P, Bisceglia C, Petracca F, Carbucicchio C, Benussi S, Maisano F, Alfieri O, Pappalardo F, Zangrillo A, Maccabelli G. Management of ventricular tachycardia in the setting of a dedicated unit for the treatment of complex ventricular arrhythmias: long-term outcome after ablation. Circulation. 2013 Apr 2;127(13):1359-68. doi: 10.1161/CIRCULATIONAHA.112.000872. Epub 2013 Feb 25. PMID 23439513
- [Background] De Luca G, Campochiaro C, Sartorelli S, Peretto G, Dagna L. Therapeutic strategies for virus-negative myocarditis: a comprehensive review. Eur J Intern Med. 2020 Jul;77:9-17. doi: 10.1016/j.ejim.2020.04.050. Epub 2020 May 10. PMID 32402564
- [Background] Wahbi K, Ben Yaou R, Gandjbakhch E, Anselme F, Gossios T, Lakdawala NK, Stalens C, Sacher F, Babuty D, Trochu JN, Moubarak G, Savvatis K, Porcher R, Laforet P, Fayssoil A, Marijon E, Stojkovic T, Behin A, Leonard-Louis S, Sole G, Labombarda F, Richard P, Metay C, Quijano-Roy S, Dabaj I, Klug D, Vantyghem MC, Chevalier P, Ambrosi P, Salort E, Sadoul N, Waintraub X, Chikhaoui K, Mabo P, Combes N, Maury P, Sellal JM, Tedrow UB, Kalman JM, Vohra J, Androulakis AFA, Zeppenfeld K, Thompson T, Barnerias C, Becane HM, Bieth E, Boccara F, Bonnet D, Bouhour F, Boule S, Brehin AC, Chapon F, Cintas P, Cuisset JM, Davy JM, De Sandre-Giovannoli A, Demurger F, Desguerre I, Dieterich K, Durigneux J, Echaniz-Laguna A, Eschalier R, Ferreiro A, Ferrer X, Francannet C, Fradin M, Gaborit B, Gay A, Hagege A, Isapof A, Jeru I, Juntas Morales R, Lagrue E, Lamblin N, Lascols O, Laugel V, Lazarus A, Leturcq F, Levy N, Magot A, Manel V, Martins R, Mayer M, Mercier S, Meune C, Michaud M, Minot-Myhie MC, Muchir A, Nadaj-Pakleza A, Pereon Y, Petiot P, Petit F, Praline J, Rollin A, Sabouraud P, Sarret C, Schaeffer S, Taithe F, Tard C, Tiffreau V, Toutain A, Vatier C, Walther-Louvier U, Eymard B, Charron P, Vigouroux C, Bonne G, Kumar S, Elliott P, Duboc D. Development and Validation of a New Risk Prediction Score for Life-Threatening Ventricular Tachyarrhythmias in Laminopathies. Circulation. 2019 Jul 23;140(4):293-302. doi: 10.1161/CIRCULATIONAHA.118.039410. Epub 2019 Jun 3. PMID 31155932
- [Background] Cadrin-Tourigny J, Bosman LP, Nozza A, Wang W, Tadros R, Bhonsale A, Bourfiss M, Fortier A, Lie OH, Saguner AM, Svensson A, Andorin A, Tichnell C, Murray B, Zeppenfeld K, van den Berg MP, Asselbergs FW, Wilde AAM, Krahn AD, Talajic M, Rivard L, Chelko S, Zimmerman SL, Kamel IR, Crosson JE, Judge DP, Yap SC, van der Heijden JF, Tandri H, Jongbloed JDH, Guertin MC, van Tintelen JP, Platonov PG, Duru F, Haugaa KH, Khairy P, Hauer RNW, Calkins H, Te Riele ASJM, James CA. A new prediction model for ventricular arrhythmias in arrhythmogenic right ventricular cardiomyopathy. Eur Heart J. 2019 Jun 14;40(23):1850-1858. doi: 10.1093/eurheartj/ehz103. PMID 30915475
- [Background] O'Mahony C, Jichi F, Pavlou M, Monserrat L, Anastasakis A, Rapezzi C, Biagini E, Gimeno JR, Limongelli G, McKenna WJ, Omar RZ, Elliott PM; Hypertrophic Cardiomyopathy Outcomes Investigators. A novel clinical risk prediction model for sudden cardiac death in hypertrophic cardiomyopathy (HCM risk-SCD). Eur Heart J. 2014 Aug 7;35(30):2010-20. doi: 10.1093/eurheartj/eht439. Epub 2013 Oct 14. PMID 24126876
- [Background] Augusto JB, Eiros R, Nakou E, Moura-Ferreira S, Treibel TA, Captur G, Akhtar MM, Protonotarios A, Gossios TD, Savvatis K, Syrris P, Mohiddin S, Moon JC, Elliott PM, Lopes LR. Dilated cardiomyopathy and arrhythmogenic left ventricular cardiomyopathy: a comprehensive genotype-imaging phenotype study. Eur Heart J Cardiovasc Imaging. 2020 Mar 1;21(3):326-336. doi: 10.1093/ehjci/jez188. PMID 31317183
- [Background] Zorzi A, Perazzolo Marra M, Rigato I, De Lazzari M, Susana A, Niero A, Pilichou K, Migliore F, Rizzo S, Giorgi B, De Conti G, Sarto P, Serratosa L, Patrizi G, De Maria E, Pelliccia A, Basso C, Schiavon M, Bauce B, Iliceto S, Thiene G, Corrado D. Nonischemic Left Ventricular Scar as a Substrate of Life-Threatening Ventricular Arrhythmias and Sudden Cardiac Death in Competitive Athletes. Circ Arrhythm Electrophysiol. 2016 Jul;9(7):e004229. doi: 10.1161/CIRCEP.116.004229. PMID 27390211
- [Background] Peretto G, Busnardo E, Ferro P, Palmisano A, Vignale D, Esposito A, De Luca G, Campochiaro C, Sartorelli S, De Gaspari M, Rizzo S, Dagna L, Basso C, Gianolli L, Della Bella P, Sala S. Clinical Applications of FDG-PET Scan in Arrhythmic Myocarditis. JACC Cardiovasc Imaging. 2022 Oct;15(10):1771-1780. doi: 10.1016/j.jcmg.2022.02.029. Epub 2022 May 11. PMID 36202457
- [Background] Peretto G, Sala S, Rizzo S, De Luca G, Campochiaro C, Sartorelli S, Benedetti G, Palmisano A, Esposito A, Tresoldi M, Thiene G, Basso C, Della Bella P. Arrhythmias in myocarditis: State of the art. Heart Rhythm. 2019 May;16(5):793-801. doi: 10.1016/j.hrthm.2018.11.024. Epub 2018 Nov 24. PMID 30476544
- [Background] Wilde AAM, Semsarian C, Marquez MF, Sepehri Shamloo A, Ackerman MJ, Ashley EA, Sternick EB, Barajas-Martinez H, Behr ER, Bezzina CR, Breckpot J, Charron P, Chockalingam P, Crotti L, Gollob MH, Lubitz S, Makita N, Ohno S, Ortiz-Genga M, Sacilotto L, Schulze-Bahr E, Shimizu W, Sotoodehnia N, Tadros R, Ware JS, Winlaw DS, Kaufman ES; Document Reviewers; Aiba T, Bollmann A, Choi JI, Dalal A, Darrieux F, Giudicessi J, Guerchicoff M, Hong K, Krahn AD, MacIntyre C, Mackall JA, Mont L, Napolitano C, Ochoa JP, Peichl P, Pereira AC, Schwartz PJ, Skinner J, Stellbrink C, Tfelt-Hansen J, Deneke T. European Heart Rhythm Association (EHRA)/Heart Rhythm Society (HRS)/Asia Pacific Heart Rhythm Society (APHRS)/Latin American Heart Rhythm Society (LAHRS) Expert Consensus Statement on the State of Genetic Testing for Cardiac Diseases. Heart Rhythm. 2022 Jul;19(7):e1-e60. doi: 10.1016/j.hrthm.2022.03.1225. Epub 2022 Apr 4. No abstract available. PMID 35390533
- [Background] Peretto G, Sala S, Basso C, Rizzo S, Radinovic A, Frontera A, Limite LR, Paglino G, Bisceglia C, De Luca G, Campochiaro C, Sartorelli S, Palmisano A, Esposito A, Busnardo E, Villatore A, Baratto F, Cireddu M, Marzi A, D'Angelo G, Gulletta S, Vergara P, De Cobelli F, Dagna L, Mazzone P, Della Bella P. Inflammation as a Predictor of Recurrent Ventricular Tachycardia After Ablation in Patients With Myocarditis. J Am Coll Cardiol. 2020 Oct 6;76(14):1644-1656. doi: 10.1016/j.jacc.2020.08.012. PMID 33004129
- [Background] Peretto G, Sala S, De Luca G, Marcolongo R, Campochiaro C, Sartorelli S, Tresoldi M, Foppoli L, Palmisano A, Esposito A, De Cobelli F, Rizzo S, Thiene G, Basso C, Dagna L, Caforio ALP, Della Bella P. Immunosuppressive Therapy and Risk Stratification of Patients With Myocarditis Presenting With Ventricular Arrhythmias. JACC Clin Electrophysiol. 2020 Oct;6(10):1221-1234. doi: 10.1016/j.jacep.2020.05.013. Epub 2020 Jun 24. PMID 33092747
- [Background] Peretto G, Mazzone P, Paglino G, Marzi A, Tsitsinakis G, Rizzo S, Basso C, Della Bella P, Sala S. Continuous Electrical Monitoring in Patients with Arrhythmic Myocarditis: Insights from a Referral Center. J Clin Med. 2021 Nov 1;10(21):5142. doi: 10.3390/jcm10215142. PMID 34768662
- [Background] Peretto G, Sala S, Rizzo S, Palmisano A, Esposito A, De Cobelli F, Campochiaro C, De Luca G, Foppoli L, Dagna L, Thiene G, Basso C, Della Bella P. Ventricular Arrhythmias in Myocarditis: Characterization and Relationships With Myocardial Inflammation. J Am Coll Cardiol. 2020 Mar 10;75(9):1046-1057. doi: 10.1016/j.jacc.2020.01.036. PMID 32138965
- [Background] Peretto G, Barzaghi F, Cicalese MP, Di Resta C, Slavich M, Benedetti S, Giangiobbe S, Rizzo S, Palmisano A, Esposito A, De Cobelli F, Gulletta S, Basso C, Casari G, Aiuti A, Della Bella P, Sala S. Immunosuppressive therapy in childhood-onset arrhythmogenic inflammatory cardiomyopathy. Pacing Clin Electrophysiol. 2021 Mar;44(3):552-556. doi: 10.1111/pace.14153. Epub 2021 Jan 18. PMID 33372694
- [Background] Asatryan B, Asimaki A, Landstrom AP, Khanji MY, Odening KE, Cooper LT, Marchlinski FE, Gelzer AR, Semsarian C, Reichlin T, Owens AT, Chahal CAA. Inflammation and Immune Response in Arrhythmogenic Cardiomyopathy: State-of-the-Art Review. Circulation. 2021 Nov 16;144(20):1646-1655. doi: 10.1161/CIRCULATIONAHA.121.055890. Epub 2021 Nov 15. PMID 34780255
- [Background] Peretto G, Sommariva E, Di Resta C, Rabino M, Villatore A, Lazzeroni D, Sala S, Pompilio G, Cooper LT. Myocardial Inflammation as a Manifestation of Genetic Cardiomyopathies: From Bedside to the Bench. Biomolecules. 2023 Apr 4;13(4):646. doi: 10.3390/biom13040646. PMID 37189393
- [Background] Ammirati E, Raimondi F, Piriou N, Sardo Infirri L, Mohiddin SA, Mazzanti A, Shenoy C, Cavallari UA, Imazio M, Aquaro GD, Olivotto I, Pedrotti P, Sekhri N, Van de Heyning CM, Broeckx G, Peretto G, Guttmann O, Dellegrottaglie S, Scatteia A, Gentile P, Merlo M, Goldberg RI, Reyentovich A, Sciamanna C, Klaassen S, Poller W, Trankle CR, Abbate A, Keren A, Horowitz-Cederboim S, Cadrin-Tourigny J, Tadros R, Annoni GA, Bonoldi E, Toquet C, Marteau L, Probst V, Trochu JN, Kissopoulou A, Grosu A, Kukavica D, Trancuccio A, Gil C, Tini G, Pedrazzini M, Torchio M, Sinagra G, Gimeno JR, Bernasconi D, Valsecchi MG, Klingel K, Adler ED, Camici PG, Cooper LT Jr. Acute Myocarditis Associated With Desmosomal Gene Variants. JACC Heart Fail. 2022 Oct;10(10):714-727. doi: 10.1016/j.jchf.2022.06.013. Epub 2022 Sep 7. PMID 36175056
- [Background] Piriou N, Marteau L, Kyndt F, Serfaty JM, Toquet C, Le Gloan L, Warin-Fresse K, Guijarro D, Le Tourneau T, Conan E, Thollet A, Probst V, Trochu JN. Familial screening in case of acute myocarditis reveals inherited arrhythmogenic left ventricular cardiomyopathies. ESC Heart Fail. 2020 Aug;7(4):1520-1533. doi: 10.1002/ehf2.12686. Epub 2020 May 1. PMID 32356610
- [Background] Lopez-Ayala JM, Pastor-Quirante F, Gonzalez-Carrillo J, Lopez-Cuenca D, Sanchez-Munoz JJ, Oliva-Sandoval MJ, Gimeno JR. Genetics of myocarditis in arrhythmogenic right ventricular dysplasia. Heart Rhythm. 2015 Apr;12(4):766-73. doi: 10.1016/j.hrthm.2015.01.001. Epub 2015 Jan 20. PMID 25616123
- [Background] Peretto G, Mazzone P. Arrhythmogenic Cardiomyopathy: One, None and a Hundred Thousand Diseases. J Pers Med. 2022 Jul 30;12(8):1256. doi: 10.3390/jpm12081256. PMID 36013207
- [Background] Peretto G, De Luca G, Villatore A, Di Resta C, Sala S, Palmisano A, Vignale D, Campochiaro C, Lazzeroni D, De Gaspari M, Rizzo S, Busnardo E, Ferro P, Gianolli L, Basso C, Dagna L, Esposito A, Benedetti S, Della Bella P. Multimodal Detection and Targeting of Biopsy-Proven Myocardial Inflammation in Genetic Cardiomyopathies: A Pilot Report. JACC Basic Transl Sci. 2023 Jul 5;8(7):755-765. doi: 10.1016/j.jacbts.2023.02.018. eCollection 2023 Jul. PMID 37547072
- [Background] Peretto G, Sala S, Della Bella P, Basso C, Cooper LT Jr. Reply: Genetic Basis for Acute Myocarditis Presenting With Ventricular Arrhythmias? J Am Coll Cardiol. 2020 Jul 7;76(1):126-128. doi: 10.1016/j.jacc.2020.05.014. No abstract available. PMID 32616153
- [Background] Peretto G, Casella M, Merlo M, Benedetti S, Rizzo S, Cappelletto C, Di Resta C, Compagnucci P, De Gaspari M, Dello Russo A, Casari G, Basso C, Sala S, Sinagra G, Della Bella P, Cooper LT Jr. Inflammation on Endomyocardial Biopsy Predicts Risk of MACE in Undefined Left Ventricular Arrhythmogenic Cardiomyopathy. JACC Clin Electrophysiol. 2023 Jul;9(7 Pt 1):951-961. doi: 10.1016/j.jacep.2022.10.032. Epub 2023 Jan 18. PMID 36752457
- [Background] Caforio ALP, Adler Y, Agostini C, Allanore Y, Anastasakis A, Arad M, Bohm M, Charron P, Elliott PM, Eriksson U, Felix SB, Garcia-Pavia P, Hachulla E, Heymans S, Imazio M, Klingel K, Marcolongo R, Matucci Cerinic M, Pantazis A, Plein S, Poli V, Rigopoulos A, Seferovic P, Shoenfeld Y, Zamorano JL, Linhart A. Diagnosis and management of myocardial involvement in systemic immune-mediated diseases: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Disease. Eur Heart J. 2017 Sep 14;38(35):2649-2662. doi: 10.1093/eurheartj/ehx321. No abstract available. PMID 28655210
- [Background] Maron BJ, Towbin JA, Thiene G, Antzelevitch C, Corrado D, Arnett D, Moss AJ, Seidman CE, Young JB; American Heart Association; Council on Clinical Cardiology, Heart Failure and Transplantation Committee; Quality of Care and Outcomes Research and Functional Genomics and Translational Biology Interdisciplinary Working Groups; Council on Epidemiology and Prevention. Contemporary definitions and classification of the cardiomyopathies: an American Heart Association Scientific Statement from the Council on Clinical Cardiology, Heart Failure and Transplantation Committee; Quality of Care and Outcomes Research and Functional Genomics and Translational Biology Interdisciplinary Working Groups; and Council on Epidemiology and Prevention. Circulation. 2006 Apr 11;113(14):1807-16. doi: 10.1161/CIRCULATIONAHA.106.174287. Epub 2006 Mar 27. PMID 16567565
- [Background] Elliott P, Andersson B, Arbustini E, Bilinska Z, Cecchi F, Charron P, Dubourg O, Kuhl U, Maisch B, McKenna WJ, Monserrat L, Pankuweit S, Rapezzi C, Seferovic P, Tavazzi L, Keren A. Classification of the cardiomyopathies: a position statement from the European Society Of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2008 Jan;29(2):270-6. doi: 10.1093/eurheartj/ehm342. Epub 2007 Oct 4. PMID 17916581
- [Background] Al-Khatib SM, Stevenson WG, Ackerman MJ, Bryant WJ, Callans DJ, Curtis AB, Deal BJ, Dickfeld T, Field ME, Fonarow GC, Gillis AM, Granger CB, Hammill SC, Hlatky MA, Joglar JA, Kay GN, Matlock DD, Myerburg RJ, Page RL. 2017 AHA/ACC/HRS guideline for management of patients with ventricular arrhythmias and the prevention of sudden cardiac death: Executive summary: A Report of the American College of Cardiology/American Heart Association Task Force on Clinical Practice Guidelines and the Heart Rhythm Society. Heart Rhythm. 2018 Oct;15(10):e190-e252. doi: 10.1016/j.hrthm.2017.10.035. Epub 2017 Oct 30. No abstract available. PMID 29097320
- [Background] Tfelt-Hansen J, Winkel BG, de Riva M, Zeppenfeld K. The '10 commandments' for the 2022 ESC Guidelines for the management of patients with ventricular arrhythmias and the prevention of sudden cardiac death. Eur Heart J. 2023 Jan 14;44(3):176-177. doi: 10.1093/eurheartj/ehac699. No abstract available. PMID 36477551